

18 January 2018

Thomas T. Henderson, MD Attn: Valerie Gatavaski, COA Eye Clinic of Austin 3410 Far West Boulevard, Suite 140 Austin, TX 78731

Re: GUARDION Health Sciences, Inc., Protocol number 1

Dear Dr. Henderson:

The Protocol Version 2 dated 27 DEC 2017, and revisions to the Informed Consent Document (ICD) were approved using the expedited review procedure on 17 January 2018, as reflected on the attached document.

Due to the nature of the modifications, the reviewer has determined that reconsenting is required. Investigators must consider enrollment at their site as of the approval date listed and ensure any participants enrolled are reconsented at the next study visit.

If you have questions, or if we can provide further assistance, please contact our office at (512) 380-1244 or at salus@salusirb.com.

Sincerely,

Trina Anderson, CCRP, CIP Quality Systems Manager

rina underson

## MODIFICATIONS TO PREVIOUSLY APPROVED RESEARCH

2111 West Braker Lane, Suite 400 • Austin, TX 78758 • P: 512.380.1244 • F: 512.382.8902 • salus@salusirb.com

| SPONSOR: GUARDION HEALTH SCIENCES | PROTOCOL #: 1 |
|---|---|
| A. INVESTIGATOR AND STUDY INFORMATION: | |
| Name of Person Completing Form: | Thomas T. Henderson, MD |
| Phone Number of Person Completing Form: | 512-427-1100 |
| Email of Person Completing Form: | thenderson@eyeclinic2020.com<br>vgatavaski@eyeclinicof austin.com |
| 4. Investigator Name: Thomas Henderson, MD OR All Investigators currently approved (multi-site s | |
| B. REQUEST FOR REVIEW/APPROVAL (Check all that a Protocol Amendment/Revision version and date: Include a detailed summary of changes/marked of Include copy of final protocol amendment or revision to the changes to the protocol require modifications of the final protocol require modifications of the second protocol require modifications of the protocol require modifications noted that the protocol require modifications noted that the protocol require modifications noted that the protocol require modifications are also please attach a rationale for modifications noted that the protocol require modifications noted that the protocol require modifications are also please attach a rationale for modifications noted that the protocol require modifications are also please attach a rationale for modifications noted that the protocol require modifications are also please attach a rationale for modifications noted that the protocol require modifications are also please attach a rationale for modifications noted that the protocol require modifications noted the protocol require modifications noted that the protocol require modification is noted to the protocol require modification is noted to the protocol requ | VUSIN 2 dated 27Dic 2017 (The sopy of protocol amendment sed protocol to the approved ICD? No Yes |
| Planned Protocol Deviations - a prospective, intenti details on the reporting these events, see the Report Other Safety Information): Describe the planned protocol deviation: Describe how the deviation is not consistent with the Provide the rationale for the planned deviation: Provide written documentation of the Spansor's are | |
| Investigator's Brochure/Product Information (ex. packat Do the changes to the IB or Product Information required If yes, please indicate below and include the requested If no, please attach a rationale for modifications not be include a detailed summary of changes Include copy of revised Investigator's Brochure/Product Information (ex. packator) Include attached Investigator (ex. packator) Include copy of revised Investigator's Brochure/Product Information (ex. packator) Include copy of revised Investigator (ex. packator) Include copy of revised Investigator (ex. packator) Include copy of revised Investigator (ex. packator) In | e modifications to the approved ICD? No Yes in modifications at this time. Ing necessary. |
| Informed consent document (ICD) revisions Include a copy of the most current IRB-approved IC for the Microsoft Word version] or handwritten chart New additional informed consent document/addendum Please note: Please remove all formatting such as all. | CD indicating changes (tracked changes [contact our office ages are acceptable for minor revisions) adding, text boxes, comments or hidden text from the ICDs |
| request and may result in additional administrative fees | such formatting may cause a delay in the review of thi |

## MODIFICATIONS TO PREVIOUSLY APPROVED RESEARCH

| sı | PONSOR: GUARDION HEALTH SCIENCES | PROTOCOL #: 1 |
|---|---|---|
| | Recruitment and Study Material | |
| | Please forward the Microsoft Word version of each file req version (number or date) in each file. | uiring review. Include the document title and |
| | ☐ New material ☐ Revised material | |
| | Identify which items and the quantity being submitted. Proposed printed advertisement, # Script of proposed video recording, # Participant screening tool, # Survey instrument(s), # Participant education material, # Other (describe): # | Proposed web site content, # Script of proposed audio recording, # Participant Diaries, # Questionnaire(s), # |
| | Request for Salus IRB to Translate Study Documents: What documents would you like translated? Consent Forms Recruitment Material Study Materials What language would you like them translated into? Language Do you require a quote before proceeding with the translated Do you require back-translation? Yes No | uage:<br>ion? |
| | Translated Documents: • Please ensure the following is attached to this request; ☐ Affidavit or Certification of accuracy from the translate ☐ A copy of the English document translated. This must ☐ A copy of the translated document. For consent form: Microsoft Word file. | ha tha mant and a trans |
| | Other items requiring review (describe): | |

## MODIFICATIONS TO PREVIOUSLY APPROVED RESEARCH

| SPONSOR: GUARDION HEALTH SCIENCES PROTOCOL #: 1 |
|---|
| THE FOLLOWING SECTIONS ARE FOR SALUS IRB USE ONLY |
| C. REVIEW AND DETERMINATION: |
| Type of Review: |
| ☐ Deferred for Full Board Review – Reviewer Signature: |
| Reviewed Only (Identify items): Investigator's Brochure/Product Information Study Material Other |
| ☑ Approved ☑ Protocol Amendment/Revision ☐ Administrative/Clarification Letter ☐ Planned Protocol Deviations ☑ Revised ICD ☐ New ICD or Addendum ☐ Recruitment/Study Material ☐ Request for Salus IRB to Translate Study Documents ☐ Translated Documents ☐ Other |
| Approved as modified (Identify items): Revised ICD New ICD or Addendum Recruitment/Study Material Other |
| EXPEDITED REVIEWER STATEMENT AND SIGNATURE: |
| The proposed modification(s) involves no more than minimal risk and represents minor changes in previously approved research during the period for which approval was granted and meets the criteria in accordance with 21 CFR 56.110 and/or 45 CFR 46.110. A minor modification means that the change does not change the risks of the research or affect the design of the research and all added procedures involve no more than minimal risk and that all added procedures fall into categories (1)-(7) of research that can be reviewed using the expedited procedure. |
| If the ICD is modified: Is re-consenting required? ☐ No ☐ Yes, at the next study visit |
| My review of this item represents that I have no conflicting interests with the Sponsor, Investigator, or Protocol. |
| Printed name of Reviewer (Chair or Designee): Mumfaz Ahmed, MD |
| Signature of Reviewer (Chair or Designee): Humba Ahul Date: 1/17/18 |

## AN AGREEMENT TO BE IN A RESEARCH STUDY INFORMED CONSENT DOCUMENT

**Sponsor:** GUARDION HEALTH SCIENCES, Inc.

**City and State:** San Diego, California

**Protocol Number and Title:** 1, Version 2: Controlled Study of the Effect of

a Medical Food Containing All Three Carotenoids and Essential Cofactors Compared to AREDS2 on Early Macular

Degeneration

**Study Doctor:** Thomas T. Henderson, MD

**Address of Study Site:** Eye Clinic of Austin

3410 Far West Blvd, Suite 140

Austin, TX 78731

**24-Hour Telephone Number:** 512-427-1100

#### **INTRODUCTION**

You are being invited to take part in a medical research study. Before you decide to take part in this study, you should read this document. This document, called an informed consent document, explains the study. Please ask as many questions as needed so that you can decide if you want to be in the study.

To be in this research study, you cannot already be in another medical research study.

You must be honest and complete in providing your medical history. Giving false, incomplete, or misleading information about your medical history, including past and present drug use, could have very serious health consequences.

The study doctor is being paid by the Sponsor to conduct this research study.

#### **PURPOSE OF THE STUDY**

The purpose of this study is to compare the effect of treatment with Lumega  $Z^{\otimes}$ , (a medical food containing lutein, zeaxanthin and meso-zeaxanthin, as well as other components) with treatment with AREDS2. AREDS 2 is a nutrient formula used for age-related vision loss that is available over the counter and marketed by Bausch & Lomb as PreserVision® AREDS 2. Lumega Z is different than PreserVision AREDS 2 in that it is available only by prescription and contains additional vitamins, antioxidants, and micronutrients.

Patients with early signs of age-related vision loss (defined for this study as having yellow deposits in the retina and no or mild abnormality of dark adaptation) that take one of the two treatments (PreserVision AREDS 2 or Lumega Z) will be compared with those with normal dark adaptation and with the other treatment group.

#### WHAT WILL HAPPEN DURING THE STUDY

Each potential patient will undergo a screening test called AdaptDx to identify patients with normal dark adaptation and those with abnormal adaptation. AdaptDx is a machine used to test dark adaptation that involves looking into a dark field and recognizing when a light appears. All patients will receive the same exams at baseline, three months and six months (for details see listing below).

Those who are confirmed as normal dark adaptation will receive no treatment because they do not need this treatment. Those who are confirmed with a few drusen on Visucam photography and mild dark adaptation difficulty (less than or equal to 10 minutes on the AdaptDx) will receive one of two treatments below for 6 months:

- Lumega Z, a medical food, containing all 3 macular pigments, 10 mg lutein, 15 mg meso-zeaxanthin, 3mg zeaxanthin as well as essential cofactors and other antioxidants
- PreserVision AREDS 2 containing 10mg lutein, 2 mg zeaxanthin

The treatment assigned to you will be assigned by chance. You have a 2 in 3 chance of being assigned to Lumega Z or 1 in 3 chance to be assigned to PreserVision AREDS2. If positive effects are noted it is possible that the study may be extended. The tasks below are part of standard diagnostic clinical eyecare practice.

• Baseline, 3 month and 6 month examinations

Medical History
Best corrected visual acuity
Best corrected contrast sensitivity (CSV-1000)
Intraocular pressure, non dilated slit lamp exam
Dark adaptation (AdaptDx, extended exam)
Macular Pigment Optical Density (Mapcat SF)
Macular Ocular Coherence Tomography (Cirrus OCT)
Fundus Photography (Zeiss Procam)

If the Sponsor determines there is a need to extend the study, you may be asked to attend extra visits, although this is not required.

LENGTH OF THE STUDY AND NUMBER OF PARTICIPANTS EXPECTED TO TAKE PART

Approximately 90 participants, ages 60 through 80, are expected to be in this study. The study will last for six months. At any point during the study, you may choose to withdraw with absolutely no penalty or questions asked. Your withdrawal will not jeopardize your relationship with the study doctor or the study staff at his clinic.

#### **SIDE EFFECTS AND OTHER RISKS**

There are no known side effects for the nutrients to be taken for this study. Lutein, zeaxanthin and meso-zeaxanthin have been studied in several thousands of people at various doses with no reports of side effects. Additionally, leutein, zeaxanthin and meso-zeaxanthin have no known drug interactions.

You must be honest in reporting anything out of the ordinary that you may experience during the study. There is a possibility that you may experience side effects from these nutrients.

#### **UNFORESEEABLE RISKS**

As noted above, there are no known risks associated with any of the procedures in the study. However, there is always a possibility that you may experience a side effect during the study. We ask that you please tell us if you believe this to be the case so that we can properly address the issue.

#### **POSSIBLE BENEFITS OF THE STUDY**

Lutein, zeaxanthin and meso-zeaxanthin could significantly reduce your risk for developing age-related macular degeneration or may delay, halt or even reverse the progression of the disease at its very earliest stages. You may also experience improvement in visual performance by participating in this study. Even if the study does not benefit you, this study could benefit other patients in the future. You will, receive a six months supply of lutein, zeaxanthin or lutein, zeaxanthin and meso-zeaxanthin at no cost.

#### **PAYMENT FOR BEING IN THE STUDY**

You will not be paid for being in this study.

#### **ADDITIONAL COSTS**

You do not have to pay for the specific study supplements. If the examinations conducted during the study would be conducted as a part of the routine care for macular degeneration, they would be submitted to your insurance plan and you would be responsible as usual, for expenses under deductibles and copays.

#### **ALTERNATIVES TO PARTICIPATION**

There are other treatments available if you decide not to be in the study.

• You may choose to buy available supplements containing Lutein, zeaxanthin and meso-zeaxanthin.

You may choose not to take any supplements at all.

#### **RELEASE OF MEDICAL RECORDS AND PRIVACY**

Your study records will be kept private. There may be times when the study doctor will not be able to guarantee privacy, such as when your study medical records are requested by a court of law or when shared with a firm in another country that does not have privacy regulations in place. Salus IRB and accrediting agencies may inspect and copy your records, which may have your name on them. Therefore, your total privacy cannot be guaranteed. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used. The following people will have access to your study records:

- Study Doctor
- Study Monitor or Auditor
- Sponsor Company or Research Institution
- Salus IRB
- Other State or Federal Regulatory Agencies

Salus IRB has approved this study and this informed consent document. Salus IRB is a committee of scientific and non-scientific individuals who review, require modifications to, and approve or disapprove research studies by following the federal laws. This group is also required by the federal regulations to provide periodic review of ongoing research studies.

#### IN CASE OF AN INJURY RELATED TO THIS RESEARCH STUDY

You must tell your study doctor if you feel that you have been injured by taking part in this study. You can tell the study doctor in person or call the number listed on the first page of this consent document. You will be treated with the same care that any other patient would receive if they suspected a side effect from treatment. No form of compensation is offered for a research related injury.

#### **LEGAL RIGHTS**

You do not lose any legal rights by signing this consent document. The above statement, "In Case of an Injury Related to This Research Study," does not stop you from seeking legal help in case of negligence.

#### **NEW FINDINGS**

During the study, you will be told of any important new findings about the nutrients used in the study. You can then decide if you still want to be in the study.

#### WHOM TO CONTACT

You may contact the study doctor or study staff at the phone number listed on the first page of this consent document:

- for answers to questions, concerns, or complaints about this research study,
- to report a research related injury, or
- for information about study procedures.

If you need medical attention please go to the nearest emergency room.

You may contact Salus IRB if you:

- would like to speak with someone unrelated to the research,
- · have questions, concerns, or complaints regarding the research study, or
- have questions about your rights as a research participant.

Salus IRB

2111 West Braker Lane, Suite 400

Austin, TX 78758

Phone: 855-300-0815 between 8:00 AM and 5:00 PM Central Time

Email: salus@salusirb.com

If you would like additional information about your rights, research in general, or IRBs, you may visit www.salusirb.com.

#### **LEAVING THE STUDY**

Taking part in this study is your choice. You may choose either to take part or not to take part in the study. You have the right to leave this study at any time. If you do not want to be in the study, there will be no penalty to you, and you will not lose any benefits to which you are otherwise entitled.

If you wish to leave this study, please call the study doctor or study staff at the telephone number listed on the first page of this consent document to schedule study exit procedures.

Your part in this study may be stopped at any time without your permission. The following people can stop your participation and/or the study itself:

- Study Doctor
- Sponsor Company
- Salus IRB
- Regulatory Agencies

If you do not follow the study procedures you may be taken out of the study.

If you withdraw from the study, no new data about you will be collected for study purposes. The study doctor will inform you whether he/she intends to either: (1) retain and analyze already collected data relating to you up to the time of your withdrawal; or (2) honor your request that your data be destroyed or excluded from any analysis.

#### **AGREEMENT TO BE IN THE STUDY**

**FOR Salus IRB USE ONLY** 

Initial draft cas: 02Nov17

This consent document contains important information to help you decide if you want to be in this study. If you have any questions that are not answered in this consent document, please ask the person explaining this document or one of the study staff.

By consenting to participate you agree that you have been given a copy of all pages of this consent document. You have had an opportunity to ask questions and received satisfactory answers to all your questions about this study. You understand that you are free to leave the study at any time without having to give a reason and without affecting your medical care. You understand that your study-related medical records may be reviewed by the company sponsoring the study and by government authorities.

### IF YOU DO NOT AGREE WITH THE STATEMENT ABOVE, YOU SHOULD NOT SIGN THIS INFORMED CONSENT DOCUMENT.

| Printed Name of Participant | |
|-------------------------------------------------------------|------|
| Signature of Participant | Date |
| Printed Name of Person Explaining Informed Consent Document | |
| Signature of Person Explaining Informed Consent Document | Date |

tla: 17Jan18

CONTROLLED STUDY OF THE EFFECT OF A MEDICAL FOOD CONTAINING

ALL THREE MACULAR CAROTENOIDS AND ESSENTIAL COFACTORS COMPARED

TO AREDS2 ON EARLY MACULAR DEGENERATION

**Sponsor:** GUARDION HEALTH SCIENCES, Inc.

15150 Avenue of Science, Suite 200

San Diego, California 92128

(800) 873-5141

Gordon Bethwaite

Vice President, Sales and Marketing

Investigator: Thomas T. Henderson, MD

3410 Far West Blvd. Suite 140

Austin, TX 78731

(512) 427-1100

Study Product: Lumega-Z Advanced Ocular Health Medical Food

**Protocol Number: 1** 

Version 2

27 DEC 2017

## Controlled Study of the Effect of a Medical Food Containing All Three Macular Carotenoids and Essential Cofactors Compared to AREDS2 on Early Macular Degeneration

#### PURPOSE:

This 6-month randomized control study is undertaken to compare the effect of treatment with LumegaZ, a medical food containing lutein, zeaxanthin, and meso-zeaxanthin, as well as essential cofactors, other antioxidants, and mitochondrial support, with the effect of treatment with AREDS2. Patients with early macular degeneration, defined as photographically visible drusen with or without abnormal dark adaptation on the AdaptDx will be randomized 2:1 and both groups will be compared to untreated patients with normal dark adaptation.

#### **BACKGROUND:**

Macular degeneration is the most common cause of blindness in people over the age of 60. The incidence of macular degeneration at all stages is 1 in 8 and is more common than diabetes and glaucoma at the same age.

The dietary carotenoids lutein and zeaxanthin (derived primarily from leafy green vegetables and other colored fruits and vegetables) as well as meso-zeaxanthin, a metabolite of lutein, are stored in the macula in all healthy retinas. This area serves central vison, and is the specific area that is affected by macular degeneration. The accumulation of these pigments results in a yellowish coloration of the retina, the concentration of which is called macular pigment density. A large multicenter trial called AREDS 2 (2013) showed that supplementing lutein and zeaxanthin reduced progression of moderate to advanced AMD by 25%. The CREST (2014) and MOST (2015) studies showed that supplementation of all 3 macular pigments resulted in normalization of the macular pigment profile and improvement in contrast sensitivity in early AMD. All 3 macular carotenoids are recognized by the FDA as 'generally regarded as safe (GRAS) for supplementation in foods.

Macular degeneration can be understood as a disease of excessive oxidation of the retinal tissue with genetic, age, dietary and light exposure components leading to accumulation of oxidized cholesterol and polyunsaturated fatty acids both on Bruch's membrane and between Bruch's membrane and the retinal pigment epithelium in a condition analogous to plaque

buildup in arteries. These deposits block transfer of waste out of the retina leading to more accumulation and block transfer of nutrients into the retina. In macular degeneration, not enough Vitamin A crosses Bruch's membrane because of the build-up, causing a localized deficiency of Retinol in the parafoveal rods. This causes slower dark adaptation after bleaching light, which is the earliest symptom of macular degeneration: difficulty driving in darkness or adapting to dark conditions increasing with aging.

Abnormal dark adaptation found by AdaptDX testing is the earliest clinical sign of macular degeneration. This has enabled diagnosis of subclinical macular degeneration with 90% positive and negative test reliability, 3-5 years before the first drusen is visible clinically. Those patients who exhibit impaired dark adaptation, whether they are subclinical with no drusen or early with mild drusen, may benefit from nutritional and /or lifestyle changes which could significantly slow the progression of the disease. This would result in maintenance of retinal health and visual performance.

It is clear that early, effective intervention in any disease process is the key to reducing morbidity. Earlier diagnosis of macular degeneration is now possible with AdaptDX testing. Effective intervention involves reducing the photo-oxidative damage of the retina caused by the visual process in the retina, and potential clearing of the early stage blockage of bidirectional transport across Bruch's membrane. Thirty percent of people over age 60 have abnormal dark adaptation. Likewise, 30% of people have an abnormal spatial profile of macular pigment indicating insufficient meso-zeaxanthin creation from lutein. Supplementing meso-zeaxanthin as well as lutein and zeaxanthin can restore the macular pigment spatial profile and improve visual performance in early macular degeneration. Early results from an as yet unpublished exploratory study in progress with such supplementation in subclinical AMD indicate improvement in MPOD and best corrected contrast sensitivity in many patients by 6 months.

A medical food is a special category of supplement approval by the FDA where physicians prescribe it for nutritional treatment of specific medical conditions. The medical food to be used by patients in this study contains not only all the macular carotenoids in micelle formulation for improved absorption, but also significant cofactors, such as vitamins, minerals, ALA, astaxanthin, N-acetylcysteine, carnosine and others. All of these ingredients working together should significantly improve the mitochondrial, antioxidant and anti-inflammatory functions of the retina. This should allow creation of less damage to critical elements of the retina and less toxic waste such as oxidized cholesterol and oxidized polyunsaturated fatty acids which are the major components of the sub-RPE and Bruch's membrane deposits. This controlled study will attempt to show that using a medical food designed to optimize retinal metabolism and antioxidant capacity will exert a positive effect in subclinical macular degeneration, which is greater than supplementation with AREDS2 and will also improve measured functions into the range of function in untreated normal patients.

#### STUDY:

All study candidates are routine patients in a general ophthalmology practice. All patients who are interested will be offered the opportunity to participate in this controlled study of the effect of a nutritional food on subclinical macular degeneration. Each patient will undergo a screening AdaptDx to separate patients with normal dark adaptation from those with abnormal dark adaptation. All patients will receive the same exams at baseline, 3 months and 6 months. For details, see the listing below. Those who are confirmed as normal with extended dark adaptation testing will receive no treatment precisely because they are defined as not having a problem needing this treatment. Those who are confirmed with early macular degeneration by photographically visible drusen and have dark adaptation scores of less than 10 minutes will receive treatment by ingesting a commercially available medical food, containing all 3 macular pigment as well as essential cofactors and other antioxidants, or AREDS2,randomized 2:1 for 6 months. If positive effects are noted, it is possible that the study might be extended. The tasks below are part of standard diagnostic clinical eyecare practice.

- Baseline, 3 month and 6 month examinations
  - History
  - Risk factors
  - Best corrected visual acuity
  - Best corrected contrast sensitivity (CSV 1000)
  - o Intraocular pressure, nondilated slit-lamp exam
  - Dark adaptation (AdaptDX, extended exam)
  - Macular pigment optical density (MapcatSF)
  - Macular ocular coherence tomography (Zeiss Cirrus OCT)
  - Fundus photography (Zeiss VisuCam Pro)

Because these patients will have additional problems found in routine clinical practice, other exams may occur for other problems and will not be considered part of the study data. Should any adverse effects be noted thought to be from the study treatment, the patient will be examined to understand the effect and if it is felt to be not significant, the patient will be asked to continue in the study. In the highly unlikely event a serious adverse effect is noted the patient will be terminated from the study and appropriate treatment will be undertaken.

#### DATA COLLECTION:

The data will be maintained on standardized forms and printable graphics, as well as in the patient's routine clinical file. To protect identifiable information, files will be locked in a file cabinet, accessible only the PI and the study coordinator. Data will be transcribed without

personally identifiable information into standard Excel files and analyzed as appropriate using standard statistical techniques.

#### STUDY REQUIREMENTS:

This study will be conducted with the protocol, good clinical practices and applicable regulatory requirements. This is a no significant risk study, using commercially available supplements, Lumega-Z or AREDS2, containing 2 or 3 of the three carotenoids that are FDA "generally recognized as safe" for food supplementation and are found in all healthy retinas. All examinations are noninvasive and are performed with FDA cleared, commercially available medical devices in routine clinical use.

The study population consists of 90 male and female patients in a routine clinical practice age 60 and over who have early macular degeneration as defined as a few drusen visible on Visucam and have an AdaptDx score less than or equal to 10 minutes. No vulnerable populations will be studied.

The patient will be studied for improvements in ocular function. Primary endpoints would be improvement in macular pigment optical density long form, improvement in best corrected contrast sensitivity and improvement in best corrected vision. Secondary endpoints would be improvement of AdaptDx long form time or a reduction in drusen.

The study supplements for each

study subject will be kept in a locked cabinet until dispensed by study staff not involved with testing to the subject.

A protocol deviation log and an adverse effect log will be kept for each subject. Immediate attention will be paid to any serious adverse events, which by the nature of the study are completely unexpected. If any injuries occur to subjects in the protocol, they are considered to be under treatment for early AMD, (diagnosis AMD, ICD H35.3131) and will be dealt with as any other medical condition or complication of treatment.

Data will be reviewed for safety and unexpected positive or negative effects after three and six month visit period are completed for all subjects.

Data will be collected in the subjects routine electronic medical record and confirmed as complete on a hard copy visit log in a study folder for each subject. Copies of each visit will be kept in the study folder. There will be a protocol deviation log, adverse events log and a study supplement log in each subjects folder.

The information collected will be used in anonymous group data analysis to be prepared for submission for potential publication. The information will not be sold or used in future research. The data can be verified through the audit trail in the subject's individual electronic medical record original source. No data will be stored on a portable device. The data will not be destroyed because it is part of medical record of care of AMD unspecified for an individual and is subject to the laws of the state of Texas and the rules of the state medical board.



2111 West Braker Lane, Suite 400 • Austin, TX 78758 • P: 512.380.1244 • F: 512.382.8902 • salus@salusirb.com

If you require assistance answering any of the questions on this form, please contact the Salus IRB at the number listed above.

| Spon | sor: Guardion Health Sciences, Inc | Protocol#: <del>LumgeaZ#</del> 1 |
|---|---|---|
| | MINISTRATIVE INFORMATION: | |
| ⊠v<br>□" | did you learn of Salus IRB? Ve are an existing client of Salus IRB Industry Publication Other: | Sponsor/CRO recommendation |
| Spor | nsor Contact Information: | |
| 1. | Name of sponsor contact: | Gordon Bethwaite |
| 2. | Sponsor name: | Guardion Health Sciences, Inc |
| 3. | Telephone: | (800) 873-5141 |
| 4. | Email: | gbethwaite@guardionhealth,com |
| Prov | ide the Primary Contact Information for IRB inquir | ies: |
| 5. | Primary contact: | ☐ Sponsor ☐ CRO ☐ Other: PI |
| 6. | Name of primary contact: | Thomas Henderson, MD |
| 7. | Name of company: | Eye Clinic of Austin |
| 8. | Name of Project Manager (PM), if different than the primary contact: | Valerie Gatavaski, COA, Study Coordinator |
| 9. | Address (including City, State and Zip): | 3410 Far West Blvd, Suite 140, Austin, TX 78731 |
| 10. | Telephone: | 512-427-1100 |
| 11. | Email: | thenderson@eyeclinicofaustin.com |
| 12. | Include name and email addresses for additional study contacts, if needed: | vgatavaski@eyeclinicofaustin.com<br>Mo Livermore, Practice Administrator<br>mlivermore@eyeclinicofaustin.com |



JT 310c+17

| Spons | sor: Guardion Health Sciences, Inc | Proto | col#: <del>LumgoaZ#</del> 1 |
|---|---|---|---|
| Provi | ide the Accounts Payable contact informa | ation OR 🗌 Check | If same as Primary Contact provided above. |
| 13. | Name of accounts payable contact: | Mo Live | rmore, Practice Administrator |
| 14. | Name of company: | Eye Clin | nic of Austin |
| 15. | Address (including City, State and Zip) | ): <b>3410 Fa</b> i | r West Blvd, Suite 140, Austin, TX 78731 |
| 16. | Telephone: | 512-427- | -1107 |
| 17. | Email:<br>(All invoices will be sent via email) | i | ore@eyeclinicofaustin.com |
| 18. | Please list any additional requirements invoicing (ex. PO numbers) | s for | |
| B. FEC | DERALLY CONDUCTED OR SUPPOR | TED RESEARCH: | : ⊠ N/A |
| 1. | Identify the department/agency supporting the research: Salus IRB currently does not review research funded by the following departments: Dept. of Defense, Dept. of Navy, Dept. of Justice, Dept. of Energy, Environmental Protection Agency | | |
| C. PRO | OTOCOL INFORMATION: | | |
| 1. | Has this research been declined to be reviewed. | | ☑ No ☐ Yes (describe in an attachment) |
| 2. | Has another IRB terminated this resear | | No ☐ Yes (describe in an attachment) |
| 3. | Protocol/study plan version and date (including any Amendments) Specify if this is a DRAFT protocol: | | Draft Protocol, LumegaZ Protocol #1, 10/15/2107 |
| 4. | If this is a DRAFT protocol, include anticipated date of submission of the FINAL protocol. | | FINAL PROTOCOL 1 10 27-2017 |
| 5. | Therapeutic area/indication: | Respiratory Hypertension Cardiovasculary Dermatology Anti-Infectives Women's Healt Urology Mental Health Other: | ☐ Neurology<br>☐ Oncology |



310c+17

| | sor. Guardion riealth Sciences, Inc Protocol #: ŁumgeaZ#1 |
|---|---|
| 6. | Data and Safety Monitoring: A system for appropriate oversight and monitoring of the conduct of the study to ensure the safety of participants and the validity and integrity of the data. Data and safety monitoring will be conducted by: □ Data Safety Monitoring Board/Committee □ Principal Investigator (PI) □ Sponsor □ Other, please attach a description □ None, please attach a rationale |
| 7. | Is the data and safety monitoring plan identified in the protocol? |
| 8. | Will you ensure the site(s) have the necessary emergency or safety equipment to conduct the study in accordance with the protocol? □ No, please explain ∨ Yes □ N/A (for minimal risk research only) |
| 9. | Will the study be posted to the ClinicalTrials.gov website? ☐ Yes ☑ No. If no, please provide a rationale: non significant risk, but will post if requested/required |
| 10. | Please list all vulnerable populations specifically targeted in this research: NONE Children Children who are wards of State Pregnant women Non-English speaking Adults who do not read and/or write |
| 11. | If any vulnerable populations have been identified, please describe the additional safeguards included in the protocol to protect the rights and welfare of these participants: |



JT 310c+17

| Spon | sor: Guardion Health Sciences, Inc Protoc | ol#: <del>LumgeaZ#</del> 1 |
|---|---|---|
| D. IN | D. INFORMED CONSENT DOCUMENT INFORMATION: | |
| 1. | ICD submitted? | ☐ No (skip to Waiver Requests section) ☑ Yes |
| 2. | Will the protocol allow the sites to use an eConsent process? If yes. This information may be found on page: | ⊠ No<br>□ Yes |
| 3. | Are there any costs to the participants? Additional costs must be disclosed in the ICD. | ☐ No<br>☑ Yes (Please describe in an attachment.) |
| 4. | Will a HIPAA Authorization be a part of the ICD? | ☐ No (skip to question 5) ☐ Yes |
| | If yes, will the authorization include permissions for future research? | <ul> <li>No</li> <li>Yes (please ensure an explanation is provided in the protocol)</li> </ul> |
| 5. | Request for a Waiver of Documentation of ICD? | No □ Yes (Please complete a waiver request) |
| WAIVER REQUESTS | | |
| 6. | Request for a Waiver or Alteration of ICD? | No □ Yes (Please complete a waiver request) |
| 7. | Request for a Waiver of HIPAA Authorization? | No □ Yes (Please complete a waiver request) |

Salusiri

310c+17 JT

| opolicor: Cuardion Health Sciences, Inc | Protocol#: LumgeeZ#1 |
|---|---|
| If you are a PM submitting for m | ulti-site research, please complete the following sections. |
| If single-site, skip to the CERTIF | ICATION AND SIGNATURE section on the following page. |
| E. DOCUMENT DISTRIBUTION Salus IRB is pleased to offer GlobeSync password-protected access to study documents. | web-portal technology to our clients providing real-time, 24-hour<br>ents, which will serve as an on-line document repository for study<br>thod for this research, Salus IRB will distribute all documents via |
| Step 1: Please provide a list of names and e documents. If you require more contacts than t separate attachment. | mail addresses of the individuals who are authorized to access study<br>the space below allows, please send additional contact information in a |
| Name | Email Address |
| Step 2: Each new user must request an accour go to <a href="www.salusirb.com">www.salusirb.com</a> , select the GlobeSync button at the to select "Request an Account", and follow the prompts to create your use | |

An email notification is sent to authorized users when study documents are available on GlobeSync. This notification will include a link to the secure site to allow access to the approved documents.

Please note: In order to ensure continued confidentiality of study documents, please notify Salus IRB of any staff changes that require us to disable GlobeSync access.

Please check here if GlobeSync™ is not feasible for you. Please provide an email address in Section A for Per Form 110B JT 310c+ 17

F. STUDY MANAGEMENT:

| 1. | Number of total sites, per the protocol: | |
|---|---|---|
| 2. | Number of sites to be submitted to Salus IRB: | |
| 3. | Describe your plan to ensure the management of information that might be relevant appropriately communicated in a timely manner to the investigative sites and Sala | ant to the protection of participants is us IRB. |
| 4. | Who will be responsible for submitting study-wide notifications or modifications in the research, such as protocol revisions/amendments, product information updates, unanticipated problems, etc., to Salus IRB? | ☐ Sponsor/Sponsor Representatives ☐ PI(s) |
| <br> | | |

FORM 100 - Initial Review (Protocol) Version: 08September2017



JT 3100+17

| | or: Guardion Health Sciences, Inc Protocol #: <del>Lung</del> | gea2 #1 |
|---|---|---|
| | If you are a PM submitting for multi-site research, please com | nolete the following sections |
| G. RE | CRUITMENT MATERIAL: | ipion die feneming scouding. |
| 1. | Will the sponsor provide template recruitment material for this research? Se the <u>Guidance on Recruitment and Study Material</u> for additional instruction. | Yes (identify below) |
| 2. | Please forward the Microsoft Word version of each file requiring review. Include the document title and version (number or date) in each file. The following template recruitment material is attached: Proposed printed advertisement, # | |
| H. STI | UDY MATERIAL: | |
| 1. | Will the sponsor provide template study material for this research? See the Guidance on Recruitment and Study Material for additional instruction. | ☑ No (skip to section I) ☐ Yes (identify below) |
| 2. | Please forward the Microsoft Word version of each file requiring review. Include the document title and version (number or date) in each file. The following study material is attached: Participant diaries, # Survey instrument(s) or questionnaire(s), # Participant education material, # Additional material to be distributed to participants (e.g. non cash gifts for long-term retention), # | |
| I. TRA | NSLATION REQUESTS: | |
| 1. | Will the documents(s) require translation? | ☐ No (skip this section)☐ Yes |
| 2. | Who will translate these documents? | Salus IRB (complete #3) Sponsor or site (skip to next section) |
| 2 | What documents would you like translated? | ☐ ICDs ☐ Recruitment Material ☐ Study Materials |
| 3. | What language would you like them translated into? | Language: |
| | Do you require a quote before proceeding with the translation? Do you require back-translation? | ☐ Yes ☐ No<br>☐ Yes ☐ No |



310ct17 JT

| Sponsor: Guardion Health Sciences, Inc | Protocol #: <del>LumgeaZ #</del> 1 |
|---|---|
| CERTIFICATION STATEMENT AND SIGNATURE: | |
| Responsibilities (single-site PIs) or the Salus IRB Reporting Guidelines for Unanticipated Problems, De understand I may contact Salus IRB at any time with grant Salus IRB the authority to review and oversee | dication, and applicable Supplemental Forms is true and accurate, esearch by Salus IRB. I have reviewed the Investigator Reporting Sponsor Reporting Responsibilities (project managers), and the eviations, and Other Safety Information [Click hyperlink(s) above]. I the questions or concerns about determinations and requirements. I the above referenced research study and certify that the study will protocol and ICD. Further, I understand that only the Salus is |
| Thomas Henderson, MD | |
| Printed Name of Principal Investigator or Project Mana | ager |
| Signature Hudusund | 10/26/17<br>Date |
| LIST OF ATTACHMENTS: | |
| REQUIRED DOCUMENTS: | |
| An electronic version (MS Word) of the proposed in the current protocol (and any Amendments). The completion of the appropriate Supplemental Form FORM 100.A - Supplemental for Drug Resear FORM 100.B - Supplemental for Device Resear FORM 100.C Supplemental for Expedited Resear FORM 100.D Supplemental for Exempt Resear FORM 100.E Supplemental for International Research | is, as appropriate.<br>ch<br>arch<br>view of Minimal Risk Research<br>arch<br>Research |
| For Recruitment and Study Material: Please forward the document title and version (number or date) in All proposed study material (diaries, survey instrur All proposed recruitment material (audio/video scri | ments or questionnaires) |

## Salusire

#### SUPPLEMENTAL FOR DRUG RESEARCH

| | Sciences Inc. | JT 310c+17 | J |
|---|---|---|---|
| Spon | Sponsor: Guardion Health Protocol #: <del>LumegaZ protesel</del> 1 | | |
| For s | tudies using two or more drugs, provide this form | for <u>each</u> <u>drug</u> : | ð |
| 1. | Is this a "first in human" use? | No ☐ Yes (first or no human data is available) | ا<br>ا |
| 2. | What is the phase of this study? | ☐ Phase I ☐ Phase II ☐ Phase III ☐ Phase IV ☒ Other: supplement | 1000 |
| 3. | Drug Name: | LumegaZ | , <u>o</u> |
| 4. | To what class does this drug belong? | medical food Or Radio-labeled (See additional submission requirements below) | るたち |
| 5. | Is this study being conducted under an IND? | <ul> <li>☐ Yes (proceed to question 6)</li> <li>OR</li> <li>☑ No, this study is exempt from the requirement of an IND, as described in 21 CFR 312.2(b)</li> <li>☐ Attach exemption category rationale and proceed to question 9.</li> </ul> | Supplemen |
| 6. | Drug IND # | # or Pending; Date the application was submitted to the FDA: | Ŋ |
| 7. | Who holds this IND? | ☐ Sponsor ☐ Investigator - If the Investigator holds the IND, please provide a written assurance (unless documented in the protocol) signed by the Investigator, that the Investigator will conduct the research as both the Sponsor and the Investigator, in compliance with the Sponsor and Investigator regulations in 21 CFR 312, in addition to 21 CFR 50, 56. | The state of the s |
| 8. | Verification of the IND is supported by (the IB may not be used to verify the IND#): | ☐ Sponsor's protocol imprinted with the IND # ☐ Written communication from the Sponsor or FDA indicating the IND # (attached) | |
| 9. | Investigator's Brochure or equivalent included? | ☐ No<br>☐ Yes - Version and Date: | |
| 10. | Is the study drug formulation approved by the FDA? If yes, please attach the product information, PDR, etc. | ☐ No<br>☑ Yes<br>Version and Date (if appl.): ( ULL VEC 270c | +17 |

Will females be excluded from participating in this study?  $\square$  Yes  $\boxtimes$  No **if yes,** please attach a medical/scientific rationale for this exclusion.

J 310c+ 1



#### SUPPLEMENTAL FOR DRUG RESEARCH

| LI | ST OF ATTACHMENTS: |
|---|---|
| F | REQUIRED DOCUMENTS: |
| | For Investigational DRUG studies only: Investigator's Brochure (or equivalent Safety Information). For DRUG studies using approved drugs: The current Package Insert (for each approved drug used in this study) For ALL studies with an IND: Documentation from the Sponsor or the FDA that verifies the IND number (the protocol may serve as documentation if the protocol is imprinted with the IND #) Attached explanation for ALL questions where a rationale or description is indicated. |
| [ | For Radio-labeled research: Radiation Safety Committee (RSC) approval letter OR Dosimetry report showing that the anticipated human radiation dose will be below the FDA maximum exposure level. |
| | <ul> <li>Include estimated millirem exposure.</li> <li>If the letter does not include dosimetry, please ensure the information is provided in another document, such as the protocol.</li> </ul> |

## SUPPLEMENTAL FOR EXPEDITED REVIEW OF MINIMAL RISK RESEARCH

Sciences Inc.

Sponsor: Guardion Health Protocol #: LumegaZ protocol 1

JT 3000+17

Name of Principal Investigator or Project Manager: Thomas Henderson, MD, principal investigator

This form must be submitted in addition to the appropriate submission forms for Initial Review.

Certain types of research may be reviewed and approved through an expedited review process. A primary criterion is that the research be of minimal risk only. Minimal risk is defined as the probability and magnitude of harm or discomfort anticipated in the research are not in and of themselves greater than those ordinarily encountered in daily life or during the performance of routine physical or psychological examinations or tests. Additionally, the purpose of the research must fit within a series of categories as stipulated by FDA (21 CFR 56.110) and DHHS regulations (45 CFR 46.110).

| Δ | ΔP | PI | IC. | ΔR | 11 | ITY: |
|---|----|----|-----|----|----|------|

| To determine whether a research project qualifies for expedited review, the protocol must indicate the | at the |
|---|---|
| research activities fulfill requirements A and B, and one of the categories outlined under C. For a proto | col to |
| be considered for expedited review, please check A and B and the appropriate category under C. | |

- A. The research activity poses no greater than minimal risk; and
- B. The identification of the subjects and/or their responses would not reasonably place the subject at risk of criminal or civil liability or be damaging to the subject's financial standing, employability, insurability, reputation, or be stigmatizing, unless reasonable and appropriate protections will be implemented so that risk related to invasion of privacy and breach of confidentiality are no greater than minimal; and
- ☑ C. The research falls under one or more of the expedited categories below. Please check all that apply.
- ☐ Category 1. Clinical studies of drugs and medical devices only when condition (a) or (b) is met.
  - (a) Research on drugs for which an investigational new drug application (21 CFR 312) is <u>not</u> required. (Note: Research on marketed drugs that significantly increases the risks or decreases the acceptability of the risks associated with the use of the product is not eligible for expedited review.)
  - (b) Research on medical devices for which (i) an investigational device exemption (21 CFR 812) is not required; or (ii) the medical device is cleared/approved for marketing and the medical device is being used in accordance with its cleared/approved labeling.
- Category 2. Collection of blood samples by finger stick, heel stick, ear stick or venipuncture as follows:
  - (a) From healthy, non-pregnant adults who weigh at least 110 pounds. For these subjects, the amounts drawn may not exceed 550 ml in an 8-week period AND collection may not occur more frequently than 2 times per week; or
  - (b) From other adults and children considering the age, weight, and health of the subjects, the collection procedure, the amount of blood to be collected, and the frequency with which it will be collected. For these subjects, the amount drawn may not exceed the lesser of 50 ml or 3 ml per kg in an 8-week period AND collection may not occur more frequently than 2 times per week.

# Guardion Health Sciences Inc. Thomas Henderson, MD Supplemental For Ex

JT 3000+17

#### SUPPLEMENTAL FOR EXPEDITED REVIEW OF MINIMAL RISK RESEARCH

| Category 3. Prospective collection of biological specimens for research purposes by noninvasive means. |
|---|
| Examples: (a) hair and nail clippings in a nondisfiguring manner; (b) deciduous teeth at time of exfoliation or if routine patient care indicates a need for extraction; (c) permanent teeth if routine patient care indicates a need for extraction; (d) excreta and external secretions (including sweat); (e) uncannulated saliva collected either in an unstimulated fashion or stimulated by chewing gum base or wax or by applying a dilute citric solution to the tongue; (f) placenta removed at delivery; (g) amniotic fluid obtained at the time of rupture of the membrane prior to or during labor; (h) supra- and subgingival dental plaque and calculus, provided the collection procedure is not more invasive than routine prophylactic techniques; (i) mucosal and skin cells collected by buccal scraping or swab, skin swab, or mouth washings; (j) sputum collected after saline mist nebulization. |
| Category 4. Collection of data through noninvasive procedures (not involving a general anesthesia or sedation) routinely employed in clinical practice, excluding procedures involving x-rays or microwaves. Where medical devices are employed, they must be cleared/approved for marketing. (Studies intended to evaluate the safety and effectiveness of the medical device are not generally eligible for expedited review, including studies of cleared medical devices for new indications.) |
| Examples: (a) physical sensors that are applied either to the surface of the body or at a distance and do not involve nput of significant amounts of energy into the subject or an invasion of the subjects' privacy; (b) weighing or testing sensory acuity; (c) magnetic resonance imaging; (d) electrocardiography, electroencephalography, thermography, detection of naturally occurring radioactivity, electroretinography, ultrasound, diagnostic infrared imaging, Doppler blood flow, and echocardiography; (e) moderate exercise, muscular strength testing, body composition assessment, and flexibility testing where appropriate given the age, weight, and health of the individual. |
| Category 5. Research involving materials (data, documents, records, or specimens) that have been collected or will be collected solely for non-research purposes (such as medical treatment or diagnosis). (NOTE: Some research in this category may be exempt from the HHS regulations for the protection of human subjects 45 CFR 46.101(b)(4). This listing refers only to research that is not exempt. |
| Category 6. Collection of data from voice, video, digital, or image recordings made for research purposes. |
| Category 7. Research on individual or group characteristics or behavior (including, but not limited to, research on perception, cognition, motivation, identity, language, communication, cultural beliefs or practices, and social behavior) or research employing survey, interview, oral history, focus group, program evaluation, human factors evaluation, or quality assurance methodologies. (NOTE: Some research in this category may be exempt from HHS regulations for the protection of human subjects 45 CFR 46.101(b)(2) and (b)(3). This listing refers only to research that is not exempt. |



#### INVESTIGATOR AND SITE INFORMATION

2111 West Braker Lane, Suite 400 ● Austin, TX 78758 ● P: 512.380.1244 ● F: 512.382.8902 ● <u>salus@salusirb.com</u>

FORM 110.A will be saved in our Investigator files for future reference. Please notify Salus IRB of any changes to the information supplied here as soon as it becomes known to the site/Investigator (PI). If you require assistance answering any of the questions on this form, please contact the Salus IRB at the number listed above.

| INIVI | INVESTIGATOR, TI | |
|---|---|---|
| IIIAAI | INVESTIGATOR: Thomas Henderson, MD | |
| 11 | TE CONTACT (for IRB inquiries): | |
| 1. | Primary contact name: | Thoma Henderson, MD |
| 2. | Research site name: | Eye Clinic of Austin |
| 3. | Phone number: | 512-427-1100 |
| 4. | E-mail (please include email addresses for additional study contacts, as needed): | thenderson@eyeclinic2020.com<br>vgatavaski@eyeclinicofaustin.com<br>mlivermore@eyeclinicofaustin.com |
| B. PR | IMARY RESEARCH SITE INFORMATION: | |
| 1. | Name of research site (Site 1): | Eye Clinic of Austin |
| 2. | Site address (including City, State and Zip): | 3410 Far West Blvd, Suite 140, Austin,TX 78731 |
| 3. | Site 24 hour phone number for participants: | 512-427-1100 |
| 4. | Pl's direct phone number for board inquiries: | 512-422-2903 |
| 5. | Pl's email: | thenderson@eyeclinic2020.com |
| 6. | For Drug or Device Research: Check all emergence life threatening allergic reactions: Anaphylactic Shock Kit CPR Trained Personnel Full Crash Cart Other (describe): | cy or safety equipment currently available at this site to treat |
| Provid | DITIONAL RESEARCH SITES OR N/A OF NONE: | by place other than the main site such as hospitals, clinics or private |
| 1. | Name of Site 2: | it could be listed in box 3 of Form FDA 1572, if applicable). |
| 2. | Complete Address (including City, State and Zip): | |
| | For Drug or Device Research: Check all emergency or safety equipment currently available at this site to treat life threatening allergic reactions: | |
| 3. | ☐ Anaphylactic Shock Kit ☐ CPR Trained Personnel ☐ Full Crash Cart ☐ Other (describe): | |
| | For Pls with more than 2 sites, please provide | the additional site information in an attachment. |
| 4. | Number of additional sites being submitted in attachr | ment, if applicable: |





| INV | INVESTIGATOR: Thomas Henderson, MD | |
|---|---|---|
| D. P | D. PRINCIPAL INVESTIGATOR CREDENTIALS AND RESOURCES | |
| 1. | The following documents must be included with this submission: | <ul> <li>☐ The PI's current professional license</li> <li>☑ already on file</li> <li>☐ The PI's current CV</li> <li>☑ already on file</li> <li>☐ PET-abc Records. Please list email address used to access these records:</li> </ul> |
| 2. | For DRUG studies taking place in Massachusetts, include: MA Researcher license already on file DEA license (controlled substance) already on file | |
| 3. | Is there any pending disciplinary action against licensing board? | the PI from ANY state No Yes (attached) |
| 4. | Describe the PI's process for ensuring that all persons assisting with the research are adequately information | |
| 5. | Describe the setting in which the research activity wind Clinical ophthalmology office | |
| 6. | Privacy refers to persons and their interest in controlling the access of others to themselves. Describe the plan to protect the privacy of research participants, during and after their involvement in the research. Participants consented away from the public areas Study-related assessments conducted in a private area Participant information collected is limited to study requirements Additional provisions (describe): locked files | |
| 7. | If no was indicated on any of the first 3 responses above, please provide an explanation: uses routine clinical examination techniques to obtain data, doors closed | |
| 8. | Confidentiality refers to the agreement between the PI and participant in how the participant's identifiable private information will be managed and used. Describe the plan to maintain the confidentiality of the data collected during and after the research is complete (check all that apply) Paper files will be kept in a secure location with limited access by authorized study staff Electronic files are password-protected with limited access by authorized study staff Participant's identifying information will be protected from improper use and disclosure (e.g. coding, making data anonymous) Research staff sign confidentiality agreements before engaging in research activities The site will not use the collected information outside of that specifically consented to and authorized Other (describe): | |



#### **INVESTIGATOR AND SITE INFORMATION**

| INV | INVESTIGATOR: Thomas Henderson, MD | |
|---|---|---|
| E. PI | E. PI EXPERIENCE AND TRAINING: | |
| uici | the PI's responsibility to ensure that all research staff assisting in the conduct robligations in meeting the requirements of 21 CFR Parts 50, 56 and 45 Cocation to follow the requirements. | of this research are informed about<br>FR 46, and have the training and |
| 1. | Has the PI completed human subject protection training? | <ul><li>☐ No</li><li>☐ Yes, attached</li><li>☒ Yes, already on file</li></ul> |
| 2. | Do any other members of the PI's staff, including Sub-Investigators, have any human subject protections training? | ☐ No ☐ Yes |
| 3. | How many years has the PI been conducting research? | 35 |
| F. RE | GULATORY INSPECTIONS: | |
| 1. | Are there any pending or active legal, regulatory, or professional actions o restrictions related to the practice of medicine or research at the site? | Yes, attached |
| 2. | Has the PI or any members of the research staff been disciplined or restricted by the FDA, DHHS or other regulatory agencies? | Yes, attached |
| 3. | Has the PI been subject to an FDA, DHHS or other regulatory agency inspection within the past 2 years? If yes, please provide inspection findings and site response or written notification from the agency. | No Yes, attached Yes, already on file |
| 4. | Has the PI been debarred by the FDA, DHHS or other regulatory agency? | <ul><li>No</li><li>Yes, attached</li></ul> |
| | FORMED CONSENT DOCUMENT (ICD) INFORMATION or N/A: | |
| Attac<br>belo<br>OR | Complete this section for consenting procedures (for all participants) at your site. OR Attach your site specific SOP regarding the consent process. If submitting a SOP, please complete the questions below for any items not addressed in your SOP. | |
| 1. | Who will present the ICD to the potential research participant and conduct the consent interview at this site? □ PI □ Sub Investigator □ Research Coordinator/ □ Other: | /Research Nurse |
| 2. | What steps will you take to minimize the possibility of coercion or undue influence? | |
| 3. | Will prospective participants be allowed to take the ICD home to discuss | Yes No (please explain in attachment) |
| 4. | Describe the timeframe between approaching the prospective participants and Timeframe may vary from a few days to a few weeks depending on the avistudy appointments | ailability of the subject and |
| 5. | Describe who will assist the PI in ensuring informed consent is appropriately obensuring that a copy is provided to the participant: research coordinator | tained and documented and for |





INVESTIGATOR: Thomas Henderson, MD

#### INVESTIGATOR STATEMENT OF AGREEMENT:

As the PI, I accept full responsibility for:

- Reviewing the protocol (and Investigator's Brochure, if applicable) in its entirety, and conducting the
  research according to the Salus IRB approved protocol. Ensuring that all research staff complies with the
  requirements of the protocol.
- Ensuring adequate and reliable financial and/or other resources are available to conduct research and halt research procedures should any of these resources become unavailable.
- 3. Ensuring that I and all research staff assisting in the conduct of research are informed about their obligations in meeting the requirements of 21 CFR Parts 50, 56 and/or 45 CFR 46, and ICH-GCP 4.1-4.13 as applicable and have the training and education to follow the requirements. Ensuring consideration of all applicable federal regulations, local and/or state laws pertinent to the research site, and consideration of community attitudes in terms of religious, ethnic, or economic status of the community from which research subjects will be drawn, relative to research at my site.
- 4. Ensuring that no member of the study staff (or their immediate family's), including sub-Investigators, has an actual or perceived Conflicts of Interest (COI) with any study, and if one is present that it will be effectively managed so to not interfere with the study progression and data.
- 5. Providing a copy of the Salus IRB approved ICD to research participants at the time of consent, and for not enrolling any individual into research until voluntary consent has been appropriately obtained and documented. Ensuring that each potential subject is provided with the information needed to understand the nature and potential risks of the research, and for taking necessary steps for the individual to gain that comprehension.
- 6. Ensuring that no individual is recruited into research: (a) until the study has been approved in writing by Salus IRB; (b) during any period wherein Salus IRB approval of a research study has lapsed; (c) during any period wherein Salus IRB approval of research or participant enrollment has been suspended, or wherein the sponsor has suspended research study enrollment; (d) following termination of Salus IRB approval of research; or (e) following expiration of the approval period as established by Salus IRB.
- 7. Promptly assessing and reporting all unanticipated problems to Salus IRB within the required timeframe, and ensuring that participants who have suffered an unanticipated problem or adverse event associated with research participation receive adequate care to correct or alleviate the consequences of the event to the extent possible. Arranging for the treatment of a research related injury with the sponsor, when applicable.
- 8. Promptly reporting all proposed changes in previously approved research to Salus IRB. Making no changes in approved research except when necessary to eliminate an apparent immediate hazard to research participants. Making no changes to the information provided to research participants (potential or active), such as ICD, recruitment or study material in electronic or print format. Promptly reporting any changes in the Pl's address or other contact information and seeking approval for an additional research facility prior to initiation of study procedures at that facility. Promptly reporting any changes to the Financial Disclosure/COI information that was initially disclosed; or occurrences of undue influence.
- 9. Ensuring that research participants are kept fully informed of any new information that may affect their willingness to continue participation in the research. For responding appropriately and adequately to all inquiries, complaints, or concerns from research participants. Promptly reporting any changes to the participant population, or in the vulnerability of participants to Salus IRB.





INVESTIGATOR: Thomas Henderson, MD

- 10. Maintaining each participant's information in such a way as to protect the privacy of the individual and the confidentiality of the data.
- 11. Seeking timely review and approval for continuing the research in accordance with 21 CFR 56.109(f) or 45 CFR 46.109(e), prior to the expiration date to avoid non-compliance with Salus IRB policies or administrative closure of the research. Notifying Salus IRB upon completion of the research and promptly submitting a

| Final/Closeout Report, as it applies to my research, prior to the expiration date of the approval period. Responding promptly to all requests for information or materials from Salus IRB board members or staff. |
|---|
| 12. For research involving investigational products (IP) (drugs/devices): Administering the IP only to participants under my supervision or the supervision of my designee(s). Supplying the IP only to those individuals who are authorized to receive it. |
| 13. I understand that <b>Finder's fees</b> (referral fees) provided by the PI/sponsor to research staff or other Physicians for potential participant referrals are not allowed by Salus IRB. Salus IRB will allow the sponsor or PI to pay a referral fee to a research participant for referring another research participant and some stipulations may apply. I further understand that <b>Recruitment bonuses</b> (payments from the sponsor to an PI or organization designed to accelerate recruitment based on the rate or timing of participant enrollment) should be disclosed to Salus IRB and will be considered by Salus IRB on a case-by-case basis. |
| My signature below indicates that; I agree to assume the responsibilities for the safe and ethical conduct of research and to abide by the decisions and requirements of Salus IRB; I have reviewed the Investigator Reporting Responsibilities and the Reporting Guidelines for Unanticipated Problems, Deviations, and Other Safety Information. [Click hyperlink(s) above]; If study staff/Sub-Investigators are permitted to sign research documents in lieu of the PI, I understand it is my responsibility to ensure that the delegated staff are notified of the reporting requirements; I may contact Salus IRB at any time with questions or concerns about these requirements; The information provided on this document is true and accurate to the best of my knowledge; to notify Salus IRB if any of the information contained in this form should |
| Signature of Principal Investigator: 14udus-WT Date: 1024/15 |
| LIST OF ATTACHMENTS: |
| REQUIRED DOCUMENTS: |
| Once the following information is submitted to Salus IRB, it will be saved in the Investigator file for future reference The Pl's current professional license The Pl's current CV Documentation of GCP training for Pl Attached explanation for any question answered "Yes" that requires an attachment |
| ADDITIONAL REQUIRED DOCUMENTS FOR DRUG STUDIES CONDUCTED IN MASSACHUSETTES: Unless already on file, current DEA License (Controlled Substance Registration Certificate) AND Researcher License. |

| LIST OF ATTACHMENTS: | |
|---|---|
| REQUIRED DOCUMENTS: | |
| Once the following informative reference The Pl's current profession The Pl's current CV Documentation of GCP tra Attached explanation for | tion is submitted to Salus IRB, it will be saved in the Investigator file for future nal license ining for PI any question answered "Yes" that requires an attachment |
| ADDITIONAL REQUIRED DO | OCUMENTS FOR DRUG STUDIES CONDUCTED IN MASSACHUSETTES: ent DEA License (Controlled Substance Registration Certificate) AND Researcher |



## PROTOCOL SPECIFIC INVESTIGATOR AND SITE RESOURCES

2111 West Braker Lane, Suite 400 • Austin, TX 78758 • P: 512.380.1244 • F: 512.382.8902 • salus@salusirb.com

If you require assistance answering any of the questions on this form, please contact the Salus IRB at the number listed above.

#### Sciences Inc.

SPONSOR: Guardion Health PROTOCOL #: LumegaZ Protocol 1

INVESTIGATOR: Thomas Henderson, MD 310c+17

A. SITE CONTACT for IRB inquiries:

| 1. | Primary contact name: | Thomas Henderson, MD |
|---|---|---|
| 2. | Research site name: | Eye Clinic of Austin |
| 3. | Phone number: | 512-427-1100 |
| 4. | Email (please include email for additional study contacts, as needed): | thenderson@eyeclinic2020.com<br>vgatavaski@eyeclinicofaustin.com<br>mlivermore@eyeclinicofaustin.com |

#### **B. DOCUMENT DISTRIBUTION**

Salus IRB is pleased to offer GlobeSync web-portal technology to our clients providing real-time, 24-hour password-protected access to study documents which will serve as an on-line document repository for study duration. If selected as the distribution method for this research, Salus IRB will distribute all documents via GlobeSync.

<u>Step 1</u>: Please provide a list of names and email addresses of the individuals who are authorized to access. If you require more contacts than the space below allows, please send additional contact information in a separate attachment.

| Name | Email Address |
|------|---------------|
| | <u> </u> |

Step 2: Each new user must request an account and create a username and password. To request an account:

- go to www.salusirb.com,
- select the GlobeSync button at the top of the screen,
- · select "Request an Account", and
- follow the prompts to create your user information.

An email notification is sent to authorized users when study documents are available on GlobeSync. This notification will include a link to the secure site to allow access to the approved documents.

Please note. In order to ensure continued confidentiality of study documents, please notify Salus IRB of any staff changes that require us to disable GlobeSync access.

Please check here if use of GlobeSync is not feasible for you. Please provide an email address in Section A for document distribution.

#### C. REGULATORY AGENCY:

## Salus III

#### PROTOCOL SPECIFIC INVESTIGATOR AND SITE RESOURCES

| 1. | If the research is federally funded or supported, OR the research will be conducted under your institution's FWA, please supply the following information: | 2) thorization form found == 4 = 0 = 1 + mm = 1 + 1 + 1 |
|---|---|---|
|---|---|---|

Guardion Health Sciences Inc.

Thomas Henderson, MD Protocol #: 1

JT 310c+17

Blank

Sciences

## PROTOCOL SPECIFIC INVESTIGATOR AND SITE RESOURCES

SPONSOR: Guardion Health PROTOCOL #: -LumegaZ Protocol 1 INVESTIGATOR: Thomas Henderson, MD 3100+17 D. RESEARCH SITE INFORMATION (as compared to FORM 110.A Investigator and Site Information): All sites where research procedures will be performed must receive IRB approval and should be listed on the site specific informed consent document (ICD) All sites identified on Form 110.A will be used for this research; Only the following site(s) identified on Form 110.A will be used for this research; Site name(s) -In addition to those site(s) identified on Form 110.A, the following site(s) not previously identified will be used for this research. Please complete Question A below. [If the following site(s) will be used for research in the future, please consider submitting an updated Form 110.A] None of the site(s) identified on Form 110.A will be used for this research. Please complete Question A below. [If the following site(s) will be used for other research in the future, please consider submitting an 1. updated Form 110,A1 A. Additional/New Site (if there is more than one (1) site, please supply this same information in an attachment): Site name(s) -Site address -24-hour number (to be listed on the ICD) -List procedures to be done at this site -E. IRB JURISDICTION: ☐ No (Please provide the Institutional Official's Is the research site(s) under the jurisdiction of a local signature below) 1. IRB (e.g., hospital, university, surgery center, or Yes (Please provide the IRB Chair's signature network)? below) N/A (Site is a private practice/clinic) Skip to section F. Institutional Official or Designee: I validate that this institution does not have an IRB and that Salus IRB may serve as the IRB of record for this research. Name of Institution: Printed Name: Title: Signature: Date: IRB Chair or Designee: I am aware that study-related procedures for the above referenced research will be conducted at our institution, and I hereby defer authority to Salus IRB to serve as the IRB of record for this research. Name of Institution: Printed Name: Title: Signature: Date:



## PROTOCOL SPECIFIC INVESTIGATOR AND SITE RESOURCES

| er | DONE OF THE PROPERTY OF THE PR |
|---|---|
| ; ; | PONSOR: Guardion Health PROTOCOL #: _LumogaZ Protecol-1 |
| like | VESTIGATOR: Thomas Henderson, MD JT 310c+17 |
| F. R | ECRUITMENT PRACTICES, MATERIAL: |
| 1. | Describe how the second of |
| 1. | patients in clinical practice asked with explanation of research if they would be willing to participate |
| | validate use of recruitment material for this research of a significant state of the same |
| 2. | Please do not submit tomplate make risk in additional instruction. No (skip to guestion #4) |
| | the sponsor/project manager (PM). |
| | Please forward the Microsoft Word version of each 51 |
| 3. | version (number or date) in each file. The following recruitment material is attached (please include quantity of each): Proposed printed advertisement, # |
| | Proposed web site content # |
| | ☐ Script of proposed video recording, # ☐ Script of proposed audio recording, # |
| | ☐ Participant screening tool # |
| | ☐ Other (describe, include quantity): |
| Res | search Participant Finder's Fees/Referral Fees: Such arrangement may place participants at risk of coercion or<br>ue influence or cause an inequitable selection of research participants. Salus ISB will |
| requ | Jests on a case-by-case basis |
| • | The payment arrangement for the referral must be approved by the board and should be disclosed in the ICD or addendum. |
| Find | der's fees paid to PIs or other physicians are never allowed. |
| 4. | Is the PI or sponsor providing a finder's fee or referral fee to participate to |
| 5. | If yes, please describe your policy regarding these fees and include the amount of the fee (or indicate if already on file with Salus IRB). |
| . ST | UDY MATERIAL: |
| | Will the site make use of study material for this research? See the Guidance on |
| 1. | Will the site make use of study material for this research? See the <u>Guidance on Recruitment and Study Material</u> for additional instruction. |
| 1. | Please do not submit template material already submitted for review by Sponsor/PM. No (skip to section H) Yes (identify below) |
| 1. | Please do not submit template material already submitted for review by Please forward the Microsoft Word version of the last |
| 1. | Please do not submit template material already submitted for review by Please forward the Microsoft Word version of the last |
| 1. | Please do not submit template material already submitted for review by Please forward the Microsoft Word version of each file requiring review. Include the document title and each): Participant diaries, # |
| | Please do not submit template material already submitted for review by No (skip to section H) Sponsor/PM. Please forward the Microsoft Word version of each file requiring review. Include the document title and each): |


| T | <u> </u> | ) <b>C</b> a |
|---|---|---|
| 11 | SPONSOR: Guardion Health PROTOCOL #: <u>LumegaZ Pretocel</u> 1 | |
| <u></u> | INVESTIGATOR: Thomas Henderson, MD \( \mathcal{J} \) 310c+ 17 | |
| H. TI | RANSLATION REQUESTS: | |
| 1. | Will the documents require translation? | <ul><li>✓ No (Go to section I)</li><li>✓ Yes</li></ul> |
| 2. | Who will translate these documents? | ☐ Salus IRB (complete #3)<br>☐ Site (skip to question 4) |
| 3. | What documents would you like translated? What language would you like them translated into | ☐ ICDs ☐ Recruitment Material ☐ Study Material |
| | Do you require a quote before proceeding with the Do you require back-translation? | translation? Language: Yes No Yes No |
| 4. | Describe your plan for recruiting and enrolling non-inot expecting to recruit | English speaking participants: |
| 5. | What language(s) do those obtaining consent speal <b>English</b> | k? |
| I. PI F | RESOURCES: | NA 51 310ct17 |
| 1. | The following documents must be included with this submission: | Form FDA 1572 (Investigational DRUG studies only) Note: Please DO NOT send original Form FDA 1572 Pl's Commitment to sponsor (For Device studies only) |
| 2. | Does the PI have access to the necessary p participants needed for this study, within the agreed | conulation and number of [7] N |
| 3. | Does the PI have the sufficient time to properly study within the agreed study period? | conduct and complete the No |
| 4. | Does the PI have an adequate number of qua facilities for the duration of the study, to conduct the | alified staff, and adequate No |
| 5. | Describe additional resources available at this site to support the conduct and account in the conduct | |
| J. PI E | EXPERIENCE AND TRAINING: | |
| 1. | Please describe any previous experience or training Macuhealth protocol 1, 35 years of experience | that the PI has which will aide in the conduct of this study: |
| 2. | Will Sub-Investigators perform procedures the PI is r licensed to perform? | not qualified and |
| 7.0 | Please describe those procedures: | |



### Sciences Inc.

| SPONSOR: Guardion Health | PROTOCOL#: LumegaZ Protoc | oL1 | |
|--------------------------------|---------------------------|-----|-----------|
| INVESTIGATOR: Thomas Henderson | , MD | IL | 31 oct 17 |

| K. RI | EQUIRED SAFETY AND EMERGENCY MEDICAL EQUIPMENT AND PSYCHOLOGICAL RESOURCES: | •• |
|---|---|---|
| 1. | Describe your plan for treating medical emergencies or providing counseling or additional psychological support that may be needed as a consequence of the research: none expected but fully equipped and trained for emergencies | |
| 2. | Do you have a written agreement with the sponsor that addresses medical care for research related injuries? This information will be disclosed in the ICD. Yes - Attach page from the contract, a statement from the sponsor, or a written explanation No - Explain your plan for addressing medical care for research related injuries | |
| 3. | Yes - Attach page from the contract, a statement from the sponsor, or a written explanation No - Explain your plan for addressing medical care for research related injuries | ex |



| · | Sciences Inc. | |
|---|---|---|
| 1 | SPONSOR: Guardion Health PROTOCOL #: LumegaZ Protocol 1 | |
| INV | ESTIGATOR: Thomas Henderson, MD JT 310c4 | - I7 |
| L. DA | TA PROTECTIONS AND CONFIDENTIALITY: | |
| 1. | Will eConsent be utilized for this research? If yes, please provide a written statement or SOP confirming the eConsent process is Part 11 compliant. | ⊠ No<br>□ Yes |
| | Sensitive Information: Information which may upset the individual being asked about the information, or that if misused, could reasonably cause discrimination or stigmatism, and result in damage to the individual's financial well-being, employability, insurability, or reputation. | |
| 2. | Will sensitive information be collected for this research? Examples include: Use or treatment for alcohol or drugs Illegal conduct or arrest record Sexual attitudes, preferences or practices Psychological or mental health information HIV or sexually transmitted diseases | ⊠ No<br>□ Yes |
| 3. | Will sensitive or individually identifiable health information, including demographic information, be collected using web-based tools, email, online surveys, etc.? | No (skip to section M) Yes |
| 2 | If yes, the website or online tool should clearly explain how the information might be used and what measures will be taken to ensure confidentiality of their data. | |
| | Attach the text version of the online tool for IRB approval. | |
| | How long will the information be stored? locked cabinet and password protected EMR | |
| | If the participant does not qualify for the research, what will happen to their data? | |
| | Will the information be stored and used in the future? If yes, please explain. | ⊠ No<br>□ Yes |
| | Will the information be sold to 3 <sup>rd</sup> parties? If yes, please explain. | ⊠ No<br>□ Yes |
| 4. | What security methods are in place to ensure protection of the sensitive information ( Replace the identifiers with a unique code and storing identifiers in a separate loc Never store identifiers on portable electronic devices, such as laptops, portable had USB memory sticks, and smart phones, unless devices are encrypted PHI will be transferred only over secure networks or as encrypted files PHI will only be transferred using encryption Remove and destroy identifiers as soon as possible De-identification: once data has been de-identified, it no longer qualifies as PHI Destruction of data. At what point will data be destroyed? permanent part of method of their data analysis will be done with de identified data | ation and/or device<br>ard drives, flash drives, |



| T-05 | Sciences Inc. |
|---|---|
| 11 | ONSOR: Guardion Health PROTOCOL #: Lumega Protect 1 |
| | /ESTIGATOR: Thomas Henderson, MD JT 310ct 17 |
| M. V | ULNERABLE POPULATIONS: |
| 1. | Please indicate all vulnerable populations that will be enrolled or may be specifically targeted for this research. IRB approval is required for the enrollment of vulnerable populations. If you decide to enroll persons from any of these categories at a later time, you may request IRB approval at that time. None Children (defined as individuals who have not reached the legal age under State Law to consent to the treatments or procedures in this research); (complete CHILDREN questions below, if applicable) Pregnant women Non-English speaking Adults who do not read and/or write (complete LAR question below, if applicable) Patients in nursing homes (complete LAR question below, if applicable) Educationally disadvantaged Economically disadvantaged Employees or family members of the PI or sponsor Students of the university or the PI participating in this research Other: |
| 2. | For each vulnerable population identified above, please provide your justification for including these populations in this study: |
| 3. | Describe the additional safeguards in place to protect the rights and welfare of these participants: |
| STU | STUDIES ENROLLING CHILDREN OR NIA (IF NOT ENROLLING): |
| 1. | In your state, what is the legal age to consent to the treatments or Age: |
| 2. | In your state, are both parents required to consent on behalf of the child? |
| 3. | Do you plan to obtain permission for children from individuals other than the No |
| 4. | If yes, other than the parents, who is legally authorized in your state to consent on behalf of a child? |
| 5. | For Drug or Device Research: Is this facility equipped to handle Pediatric emergencies? |



| I | Sciences Inc | |
|---|---|---|
| SPONSOR: Guardion Health PROTOCOL #: LumegaZ Protocol 1 | | |
| IN | INVESTIGATOR: Thomas Henderson, MD 31 Oct 17 | |
| SI | TUDIES USING LEGALLY AUTHORIZED REPRESENTATIVE (LAR); (If the ows LARs for participants other than children) OR NA (NOT LITTLE INC.) | ne research you are noticing. |
| all | OT EZ MA (NOT OTILIZING | LARS): |
| 1. | Who may serve as an LAR to provide consent for procedures performed | d in research? |
| | STATE AND LOCAL RESEARCH LAWS: | |
| COI<br>HIV<br>no | ease indicate any state or local laws regarding medical research and/or vulnduct of the study or that require additional information to be included in to VICDs, mandatory reporting of positive HIV/hepatitis results). | nerable populations that may affect the he ICD (e.g., separate state mandated |
| O. C | COMMUNITY ATTITUDES AND INFORMATION: | |
| 1. | Are there any community attitudes (including religious, other) at a large star and a second star at a second | |
| P. P. | AYMENT ARRANGEMENTS: | |
| <u> </u> | The following will be used to customize the ICD f | or your site: |
| 1. | Will participants be paid for their participation? | ⊠ No (skip to question 6) ☐ Yes |
| 2. | Please provide the breakdown (per visit/procedure) for compensation to the aution (compensation to the aution) | |
| | Approximately when should the participants expect payment? Payment at each study visit | |
| 3. | Payment at the participant's final visit | TT C. |
| Payment after the participant completes the study within the following time frame: | | |
| | Other (describe): | |
| 4. | Total potential compensation for completion of protocol requirements: | |
| 5. | Is an end of study bonus being offered to participants? Ensure the amount does not exceed 50% of the total payment for completion of the | □No |
| | 1,0000,017. | Yes (amount): |
| 6. | Is the PI receiving a "recruitment bonus" from the sponsor based on the rate or timing of enrollment? If yes, please attach a description of the financial arrangement and disclere. | 57.41- |
| | financial arrangement and disclose this information in the Conflicts of Interest (COIs) section. | ⊠ No<br>□ Yes |



Sciences Inc.

| SPONSOR: Guardion Health | PROTOCOL#: Lum | <del>ogaZ Protossi</del> 1 | |
|---|---|---|---|
| INVESTIGATOR: Thomas Henderson | MD | JT | 310ct 17 |

#### **CONFLICTS OF INTEREST:**

| the<br>res<br>fan<br>live | The PI is responsible for reading each statement thoroughly before signing this form. Please consider any potential, actual, or perceived conflicts of interest (COIs) of a financial, professional, or personal nature with the sponsor, test article, or manufacturer of the test article, that may affect any aspect of this research. The responses must also consider any COIs of the PI's immediate family members. Salus IRB defines "immediate family member" as (at a minimum) an individual's dependent children or a person with whom an individual lives, in the same residence, where both individuals share responsibility for each other's welfare and financial obligations (e.g., spouse, domestic partner). | |
|---|---|---|
| 1. | Do you have a financial arrangement with the sponsor, whereby the value of compensation could be influenced by the outcome of the research? This includes compensation that could be greater for a favorable clinical result, compensation in the form of an equity interest in the sponsor, or compensation tied to sales of the product or service being tested (e.g., royalty interest). | ⊠ No<br>□ Yes |
| 2. | Do you have a proprietary interest in the product or service being tested such as patent rights, trademark, copyright or licensing agreement? | ⊠ No<br>□ Yes |
| 3. | Do you have a significant equity interest in the sponsor or in the product or service being tested (e.g., ownership interest, stock options, or any other financial interest) the value of which cannot be readily determined through reference to public prices, any equity interest in the sponsor (if publicly traded) exceeding \$10,000 (or \$5,000 for PHS-funded research), or more than 5% ownership (or any combination of these), in the sponsoring company or business entity? | ⊠ No<br>□ Yes |
| 4. | Have you received payments from the sponsor or payments related to the product or service being tested in excess of \$10,000 (or \$5,000 for PHS-funded research), when aggregated for immediate family members, exclusive of the costs of conducting the research, such as honoraria, a grant or grants to fund ongoing research, compensation in the form of equipment, or retainers for ongoing consultation? | ⊠ No<br>□ Yes |
| 5. | Have you accepted payment arrangements from the sponsor such as financial incentives for early enrollment or high enrollment (e.g., recruitment bonus incentives)? | ⊠ No<br>□ Yes |
| 6. | Do you have any board or executive relationship to the sponsor or the product or service being tested, regardless of the compensation? | ⊠ No<br>□ Yes |
| 7. | Are you an employee of the sponsor or the manufacturer of the test article? | ⊠ No<br>□ Yes |
| 8. | Do any of the research staff or their immediate family members have financial or other COIs with the sponsor conducting this research, the test article, or the manufacturer of the test article, as listed above? Salus IRB defines "research staff" as anyone responsible for the design, conduct, or reporting of research (e.g., sub-investigators, research coordinators). | ⊠ No<br>□ Yes |
| be m | If you answered "Yes" to any of the questions above, <b>describe the COI(s) in detail</b> and explain how the COI(s) will be managed so that the conflict(s) will not adversely affect the protection of participants or the integrity of the research (notification of the existence of a COI and how it will be managed may be added to the ICD): | |



Sciences Inc.

| Partition Health | ىىك :# ROTOCOL | megaZ Protocci 1 | | |
|---|---|---|---|---|
| INVESTIGATOR: Thomas Henderson, N | ID | JI | 21/ | 0c+17 |
| CERTIFICATION STATEMENT AND SIGNA | Tilo | | 3' ' | |
| / certify that the information provided it | | | | |
| I certify that the information provided with<br>represents my intent to pursue review of thi | in this application<br>is research by Sai | is true and accurate | to the b | est of my knowledge, and |
| ☐ I have reviewed the lovesticator Com | | wy digiratare | Delow HI | |
| <ul> <li>I have reviewed the Investigator Rep<br/>Problems, Deviations, and Other Safety</li> <li>☑ If study staff/sub-investigators are perm</li> </ul> | <u>Information</u> . <i>[Clic</i> | <u>llities</u> and the <u>Repo</u><br>k hyperlink(s) above | orting Gu | idelines for Unanticipated |
| responsibility to ensure that the data | nitted to sign rese | earch documents in I | İ <del>A</del> U Of the | DI Lundomto de la |
| | ıs IRB; | probindes as a PI, ap | opiicable . | regulations, Good Clinical |
| ☐ I understand that it is my obligation to re☐ I attest that the information submitted to me on 10/26/17 is true and accurate. | view the Investiga<br>Salus IRB on Fo | tor's Statement of Ag | reement | on Form 110.A; |
| The on ADIZBIL Is true and accurate. | | rost - investige | nor and S | site information signed by |
| By signing this form, I grant Salus IRB the certify that the study will not begin until I have understand that only the Salus ISB. | authority to app | rove and oversee th | e above | referenced reserved |
| certify that the study will not begin until I have understand that only the Salus IRB-approved | received Salus<br>I ICD may be use | IRB approval of the | FINAL pro | otocol and ICD. Further, I |
| Thomas Henderson, MD | | and on on paracipant | ა. | |
| Printed Name of Investigator | | | | |
| $\mathcal{M}_{i}$ | _ | | | |
| Signature of Investigator | in | | | 18/26/10 |
| | | | | Date |
| IST OF ATTACHMENTS: | | | | |
| REQUIRED DOCUMENTS: | | | | |
| Completed and signed <i>Protocol Specific F</i> The sub-investigator's (performing proced | PI and Site Resou | Tes Form (this door | ···4) | ncontraction and a second |
| professional licence if | area rie el 18 110f | qualified and licenser | to name. | m) current CV and |
| any question | answered "Yes" | that requires an est- | iture refer | ence. |
| of Recruitment and Study Material: Please | forward the Mic | rosoft Word version | n of eac | h file roquisi |
| All proposed study material (diaries, surve | <b>per or date)</b> in ea<br>y instruments, or o | ich file.<br>Juestionnaires) | ·· O. Cac | ine requiring review. |
| All proposed recruitment material (audio/vi | deo script, print a | dvertisement) | | 100 TO AND COMP. A TO |

October 27, 2017

Salus IRB Form 100 Initial Review (Protocol)

Section D - Description

The ICD clearly states additional costs: You do not have to pay for the specific study supplements. Since these same tests would be conducted as part of the routine care for macular degeneration, they would be submitted to your insurance plan and you will be responsible as usual, for expenses under deductibles and copays.



#### Ingredients Serving Size: 0.75 FL, OZ, (1.5 Tbsp) Servings Per Container: 7 Amout Per Serving 0.75 FL, OZ. % Daily Value Calories Vitamin C (as ascorbic acid and calcium ascorbate) 500 mg 833% Vitamin D3 (as cholecalciferolin MCT) 2000 IU 500% Vitamin E (as mixed tocopherols with not less than 200 IU 665% 50 mg of gamma tocopherol) Thiamin (vitamin B1 as thiamin HCI) 1.5 mg 100% Riboflavin 1.7 mg 100% Niacin (as niacinamide) 20 mg 100% Vitamin B6 (as pyridoxine HCI) 10 mg 500% Folate (as folic acid) 800 mcg 200% Vitamin B12 (as methylcobalamin) 1000 mcg 16,667% Biotin 100 mcg 33% Pantothenic Acid (as d-calcium pantothenate) 10 mg 100% Calcium (as calcium lactate gluconate) 250 mg 25% Magnesium ( as magnesium citrate) 100 mg 25% Zinc (as zinc amino acid chelate) 25 mg 167% Selenium (as selenium sodium selenate) 70 mcg 100% Copper (as copper gluconate) 2 mg 100% Manganese (as manganese gluconate) 2 mg 100% Chromium ( as chromium picolinate) 100% 120 mcg Molybdenum (glycinate chelate) 75 mcg 100% NAC (N-acetyl-cysteine) 500 mg Acetyl-L-Carnitine 500 mg L-Taurine 500 mg Quercetin 100 mg CoQ10 (as ubiquinone) 50 mg Lutein\*\* 15 ma Meso-zeaxanthin\* 10 mg Zeaxanthin\* 3 mg Astaxanthin 1000 mcg Lycopene 500 mcg Proprietary Ocular Antioxidant Blend 200 mg (bilberry fruit extract 4:1, alpha-lipoic acid) \* Daily value not established.

Other Ingredients: Purified water, vegetable glycerin, polysorbate 80, acacia gum, soybean lecithin, malic acid, natural flavors, sucralose, potassium sorbate, sodium benzoate, medium chain triglycerides.

\*\*Contains *Nutri-Mz* and sold subject to US patents 6,218,436 and 6,329,432 and others worldwide.

NO sugar, yeast, gluten, or dairy.

#### Omega Boost

| Ingredient Facts Serving Size: 2 Soft Gels | Servings P | er Container: 30 |
|---|---|---|
| | Amout Per Serving | % Daily Value |
| Calories | 10 | |
| Calories from Fat | 10 | |
| Total Fat | 1.5 g | 2% |
| Saturated Fat | 0 g | 0% |
| Polyunsaturated Fat | 1 g | t |
| Monounsaturated Fat | 0 g | t |
| Fish Oil Concentrate | 1260 mg | † |
| DHA (docosahexaenoic acid) | 620 mg | t |
| EPA (eicosapentaenoic acid) | 160 mg | † |

**Ingredients:** Alaska Walleye Pollock (theragra chalcogramma), gelatin, glycerin, purified water, mixed natural tocopherols.

NO aluten, dairy, or artificial colors or flavors.



Each 4-week supply includes:
4 bottles x 5.25 Fl. Oz.
Lumega-Z Medical Food
With 60 Omega Boost Soft Gels



To order LUMEGA-Z, go online at: www.lumegaz.com or call (800) 873-5141



Formulated and distributed by: Guardion Health Sciences, Inc. San Diego, California



Patent Pending



The Medical Food created to restore and maintain the Macular Pigment

Contains all three macular carotenoids:

Lutein

Zeaxanthin

Meso-zeaxanthin

of critical Micronutrients and
Omega 3's

#### What is Lumega-Z?

Lumega-Z is a medical food created to restore and maintain the macular protective pigment.

Macular pigment protects the macula (the part of your retina responsible for sharp, central vision) against oxidative stress, free radicals, and damaging blue light.



Example of a depleted macular pigment



Example of a restored macular pigment

A depleted macular pigment is a known high risk factor for age-related macular degeneration and other retinal diseases.

#### What is Medical Food?

A Medical Food is not a drug. It is not a supplement either.



Medical foods are a regulated category of product "... formulated to be consumed or administered... under the supervision of a professional healthcare provider and intended for the specific dietary management of a disease or condition for which distinctive nutritional requirements, based on recognized scientific principles, are established by medical evaluation."

(Per Section 5(b) of the Orphan Drug Act)



Restores and maintains a depleted macular pigment

Decreases glare and light sensitivity

Liquid formula is easy to swallow and digest

Promotes overall ocular health

Can replace your daily multivitamin

Able to be purchased with Healthcare Flexible Spending Account (FSA)

Tax-deductible as a medical expense

All research and scientific data is available upon request.

### PreserVision AREDS 2 Formula Eye Vitamins for AMD

#### Thomas Henderson MD

Thu 10/26/2017 11:32 PM

To:Valerie Gatavaski <vgatavaski@eyeclinicofaustin.com>;

Cc:Thomas Henderson MD <thenderson@eyeclinicofaustin.com>;

Sunday, October 15, 2017 4:26 PM

### PreserVision AREDS 2 Formula

PreserVision AREDS 2 Formula builds on the original, clinically proven PreserVision AREDS Formula, with lutein and zeaxanthin replacing beta-carotene, based on the AREDS2 study.\*

**PreserVision** AREDS 2 Formula exactly matches the nutrient formula recommended by the AMD experts at the National Eye Institute based on the AREDS2 study.



| National Eye Institute Recommended Formula: | | |
|---|---|---|
| Nutrient | Amount (per day) | Percent Daily Value* |
| Vitamin C | 500 mg | 840% |
| Vitamin E | 400 IU | 1340% |

| Zinc | 80 mg | 540% |
|---|---|---|
| Copper | 2 mg | 100% |
| Lutein | 10 mg | ** |
| Zeaxanthin | 2 mg | ** |
| *Percent Daily Values ( | DV) based on a 2,000-calorie diet | |
| **Daily Value (DV) not | established | |
| Speak with your doctor | to determine if the updated AREDS | 2 formula is right for you |

**PreserVision** AREDS 2 formula exactly matches the levels of clinically proven nutrients recommended by the National Eye Institute based on the AREDS2 study.

PreserVision AREDS 2 Formula Eye Vitamins for AMD

http://www.preservision.com/products/preservision-areds-2-formula

Screen clipping taken: 10/15/2017 4:26 PM

Created with Microsoft OneNote 2016.

#### **CURRICULUM VITAE**

### Thomas T. Henderson, M.D., F.A.C.S.

Current Position: President and Chief Executive Officer

Eye Clinic of Austin, PLLC Thomas Henderson Sole Mbr

**Business Address:** Eye Clinic of Austin

3410 Far West Boulevard, Suite 140

Austin, Texas 78731

**Business Phone:** (512) 427-1100 Main

(512) 427-1207 Main Fax

Web Address / Electronic Mail: www.eyeclinic2020.com

thenderson@eyeclinic2020.com

Birthdate: January 12, 1947

Birthplace: Wichita, Kansas

Licensure & Certifications: Physician Permit, Texas F4863

June 13, 1979 to Present

Medicine & Surgery, Virginia 0101026396

December 6, 1975 to Present

American Board of Ophthalmology

Written exam, passed 98<sup>th</sup> percentile, January 1980

Oral exam, passed, October 1980
National Board of Medical Examiners

Passed, 1973

American College of Surgeons - Fellow

Certified, October 1997

Education & Internships: Medical Doctor

University of Texas

Southwestern Medical School

Dallas, Texas 1969 to 1973

Bachelor of Science, Psychology

Louisiana State University

1965 to 1969

#### **Surgery Externship**

Presbyterian Hospital Dallas, Texas 1971

#### **OB/GYN Externship**

Parkland Memorial Hospital Dallas, Texas 1972

#### **Rotating Internship**

San Francisco General Hospital Medical Center San Francisco, California 1973 to 1974

#### Residency in Ophthalmology

Baylor College of Medicine Houston, Texas 1976 to 1979

Post Graduate
Medical Experience:

#### Lieutenant Commander

U.S. Public Health Service, Commissioned Corps General Medical Officer Norfolk, Virginia 1974 to 1975 Galveston, Texas 1975 to 1976

Ophthalmology Practice Experience: Private Practice:

### Thomas Henderson, M.D., P.A., d.b.a.

**Eye Clinic of Austin** 

3410 Far West Boulevard, Suite 140 Austin, Texas 78731 December 1990 to Present 900 East 30<sup>th</sup> Street, Suite 200 Austin, Texas 78705 January 1982 to December 1990

#### **Medical Center Eye Associates**

Houston, Texas August 1980 to December 1981

#### Rugley-Blasingame Clinic

Wharton, Texas July 1979 to May 1980

### **Voluntary Clinical Faculty:**

Supervision of Resident Surgical Cases
Baylor College of Medicine
Department of Ophthalmology

Curriculum Vitae, Page 2 Thomas Henderson, M.D. 10/23/2013 Houston, Texas 1980 to 1981

#### **Hospital Affiliations:**

Northwest Hills Surgical Hospital (formerly HealthSouth)

Austin, Texas Chief of Staff, 1995 to 2003 1995 to Present

**Texan Surgery Center** 

Austin, Texas 2004 to Present

**Austin Diagnostic Clinic** 

Ambulatory Surgery Center – Lakewood Austin, Texas 2005 to Present

The Hospital at Westlake Medical Center

Austin, Texas 2006 to Present

**Academy of Laser Vision Sciences** 

Austin, Texas 2003 to Present

Seton Health Care

Brackenridge Hospital
Seton Medical Center
Seton Northwest Hospital
Dell Children's Hospital of Austin
Austin, Texas 1982 to Present

St. David's Healthcare Partnership

St. David's Medical Center\*
South Austin Hospital
Bailey Square Surgery Center 2005 to Present
Austin, Texas 1982 to Present
\*Chief of Ophthalmology 1997 to 1999
\*Chief of Operations 1988 to 1990

Previous Affiliations:

Park Plaza Hospital – Houston, Texas 1990 to 1991
Austin Surgical Center – Austin, Texas 1986 to 1995
Harris County Hospital – Houston, Texas 1980 to 1981
Twelve Oaks Hospital – Houston, Texas 1980 to 1981
Polly Ryan Memorial – Richmond, Texas 1979 to 1980
Gulf Coast Medical Ctr – Wharton, Texas 1979 to 1980
Caney Valley Memorial – Wharton, Texas 1979 to 1980

Curriculum Vitae, Page 3 Thomas Henderson, M.D. 10/23/2013

#### **Honors & Awards:**

Austin HealthCare Hero Nominee 2009
Best Doctors in America, 1996 to 2012
Texas Super Doctor, 2005, 2006, 2008, 2009, 2011 & 2012
Guide to America's Top Ophthalmologists 2006, 2009, 2010, 2011 & 2012
LaserVision's® Top 100 Surgeons 2008
Austin Top Refractive Eye Surgeons 2008
Consumers' Guide to Top Doctors 2003
Southwestern Medical School class Rank #1 in senior year, 26/105 overall

Louisiana State University - Phi Kappa Phi (National Honor Society)

#### **Professional Organizations:**

American Academy of Ophthalmology
Texas Ophthalmological Association
Austin Ophthalmological Society (1993, President)
American Society of Cataract and Refractive Surgery
International Society of Refractive Surgery of A.A.O.
American Medical Association
Texas Medical Association
Travis County Medical Society
American College of Eye Surgeons
American College of Surgeons
Contact Lens Association of Ophthalmologists

#### **Teaching Experience:**

Cedar Creek Elementary School Austin, Texas Lecturer "Dangers of Children's Ballgames" March 1982

Texas Society to Prevent Blindness Austin, Texas Public Service Representative – Two radio broadcasts July 1981

University of Houston, College of Optometry Houston, Texas Lecturer "Preventable Blindness Sub-Retinal Neo Vascular Membranes" April 1981

Ben Taub Hospital Houston, Texas Instructor – Resident Surgery/Ophthalmology 1980 to 1981

Gulf Coast Medical Center Wharton, Texas Lecturer "Sarcoid and the Eye" Clinical 1979

Curriculum Vitae, Page 4 Thomas Henderson, M.D. 10/23/2013

#### **Clinical Studies:**

Baylor College of Medicine Houston, Texas Ophthalmic Assistants Program: Instructor "Light, Form & Color" & "Optics & Refraction" 1977 to 1978

- Allergan, ISOP-101-8702, Sub-Investigator
- Ciba Giegey Protocol 19684A, Primary
- Pharmaco, RG121561, Sub-Investigator
- Organon, Birth Control, Sub-Investigator
- Insite Vision Pilasite/Pilopine, Primary
- Merck, Sharpe & Dohme MK507 Compassionate
- Pharmacia, Xalatan, Open Label
- Alcon, Timolol, Triple Masked
- Alcon, Olopatadine QD, November 2001
- Alcon, Blepharitis, Ciprodex, 2002 to 2003
- Alcon, Brimonidine Tartarte Generic 2003 to 2004
- Otsuka, Dry Eye Study 2004 to 2006 Primary
- Insite Vision, C-04-35 Allergic Conjunctivitis 2004
- Alcon, Allergic Conjunctivitis, Olopatadine 2004-05
- Novartis CASM981E2205, Dry Eye 2004-05
- Bausch & Lomb 433 Bacterial Conjunctivitis 2006
- Alcon, C-07-40 Phase 3 Blepharitis 2008-2009
- Alcon, C-08-47 Travatan-Z 2008-2009
- Inspire Pharmaceuticals, 03-113 Dry Eye 2009
- Inspire Pharmaceuticals, 044-101 Blepharitis 2009
- Alcon, C-09-034 Allergic Conjunctivitis 2010
- Fovea Pharmaceutical's Fov 1101-11 2010

#### **Continuing Education:**

- American Academy of Ophthalmology Focal Points 1995 (Reading Assignment) January 29, 1996
   Category 1, Hours: 15.0
- Presbyterian Hospital Dallas, TX
   18<sup>th</sup> Annual Spring Ophthalmology Symposium
   The Business of Success
   March 8, 1996
   Category 1, Hours: 7.0
- Texas Medical Association Austin, TX Witness for the Defendant Physician May 10, 1996

Curriculum Vitae, Page 5 Thomas Henderson, M.D. 10/23/2013

Category 1, Hours: 3.0

Texas Medical Association – Austin, TX
 Texas Ophthalmology Association Refractive
 Symposium
 May 11, 1996
 Category 1, Hours: 3.5

- Texas Medical Association Austin, TX Legislative Workshop May 11, 1996 Category 1, Hours: 2.0
- Texas Medical Association Austin, TX
   OMIC Workshop
   May 11, 1996
   Category 1, Hours: 3.0
- Baylor College of Medicine Houston, TX
   Baylor Welsh Cataract & Refractive Surgical
   Congress
   September 5 7, 1996
   Category 1, Hours: 20.0
- American Academy of Ophthalmology Chicago, IL Annual Meeting: VISX PRK Course & Lab October 25-27, 1996 through November 1997 Category 1, Hours: 16.0
- American Academy of Ophthalmology Chicago, IL Annual Meeting: Reshaping the Future: Refractive Surgery
   October 25-27, 1996
   Category 1, Hours: 12.0
- American Academy of Ophthalmology Chicago, IL 1996 Annual Meeting October 31, 1996
   Category 1, Hours: 16.0
- American Academy of Ophthalmology Focal Points 1996 (Reading Assignment) January 8, 1997 Category 1, Hours: 15.0
- Scott and White Memorial Hospital Temple, TX

Everett R. Veirs Lecture & Ophthalmology Conference February 21-22, 1997 Category 1, Hours: 8.0

- Presbyterian Hospital Dallas, TX
   19<sup>th</sup> Annual Spring Ophthalmology Symposium Resurfacing the Future March 14, 1997
   Category 1, Hours: 7.0
- American Academy of Ophthalmology and Texas Ophthalmology Association – Dallas, TX CodeQuest Ophthalmic Coding College 1997: Coding, Documentation & Compliance Seminar March 15, 1997 Category 1, Hours: 7.0
- American Society of Cataract & Refractive Surgery & American Society of Ophthalmic Administrators – Boston, MA
   Symposium on Cataract, IOL & Refractive Surgery April 26-30, 1997
   Category 1, Hours: 40.0
- St. David's Hospital Austin, TX
   St. David's Grand Rounds; Treatment for Chronic Pain Syndrome
   July 18, 1997
   Category 1, Hours: 1.0
- Presbyterian Hospital Dallas, TX
   Cataract 1997
   September 12, 1997
   Category 1, Hours: 7.0
- Barnet Dulaney Eye Foundation San Antonio, TX Advanced Concepts in Phacoemulsification September 20, 1997 Category 1, Hours: 6.5
- Barnet Dulaney Eye Foundation San Antonio, TX Refractive Update: Techniques, Technology & Results
   September 20, 1997
   Category 1, Hours: 4.5

- LaserVision Centers, Inc. Austin, TX
   Laser In-Sita Keratomileusis Fellowship Program
   LASIK Study Group
   October 11-12, 1997
- Bausch & Lomb Austin, TX
   C-LASIK Course
   October 11-12, 1997
- American College of Surgeons Chicago, IL Clinical Congress 1997
   October 12-17, 1997
   Category 1, Hours: 3.0
- American Academy of Ophthalmology –
   San Francisco, CA
   Reshaping the Future Refractive Surgery
   October 25, 1997
   Category 1, Hours: 13.0
- American Academy of Ophthalmology –
   San Francisco, CA
   Subspecialty Day 1997 Scientific Exhibits &
   Programs
   October 26, 1997
   Informal, Hours: 9.0
- American Academy of Ophthalmology -San Francisco, CA
   Current Concepts in the Management of Glaucoma October 26, 1997
   Category 1, Hours: 1.0
- American Academy of Ophthalmology Focal Points 1997 (Reading Assignment) January 12, 1998 Category 1, Hours: 15.0
- American Heart Association
   Advanced Cardiac Life Support
   March 11, 1998
- American Management Association How to Get More Organized

#### March 19, 1998

 Excerpta Medical Office of Continuing Medical Education
 Open Angle Glaucoma: A Focus on Current Management
 April 14, 1998
 Category 1, Hours: 2.0

Johns Hopkins University School of Medicine
 Office of Continuing Medical Education
 Hopkins Business of Medicine Executive Medical
 Business Certificate;
 Managed Care: Perspectives & Practices
 April 8, 1998 to June 10, 1998

Category 1, Hours: 30.0

Johns Hopkins University School of Medicine
 Office of Continuing Medical Education
 Hopkins Business of Medicine Executive Medical
 Business Certificate;
 Accounting for Decision Making in Medicine
 September 9, 1998 to November 18, 1998
 Category 1, Hours: 30.0

- Johns Hopkins University School of Medicine
   Office of Continuing Medical Education
   Hopkins Business of Medicine Executive Medical
   Business Certificate;
   Managerial Finance for Medical Services
   February 22, 1999 to April 26, 1999
   Category 1, Hours: 30.0
- St. David's Medical Center Austin, TX
   St. David's Grand Rounds; Antibiotic Update
   March 2, 1999
   Category 1, Hours: 1.0
- Johns Hopkins University School of Medicine Office of Continuing Medical Education Hopkins Business of Medicine Executive Medical Business Certificate; Leadership & Organizational Behavior in Medical Settings May 3, 1999 to July 12, 1999 Category 1, Hours: 30.0

- American Academy of Ophthalmology Refractive Subspecialty Day 1999: Scientific Exhibits & Programs October 22-23, 1999
   Informal, Hours: 9.0
- SLACK, Inc. Dallas, TX
   Selective Laser Trabeculotherapy:
   An Innovative Treatment for Glaucoma
   October 24, 1999
   Category 1, Hours: 2.5
- The Barnet Dulaney Eye Foundation –
   San Antonio, TX
   Advanced Concepts in Cataract & Refractive
   Surgeries
   September 9, 2000
   Category 1, Hours: 7.0
- The Barnet Dulaney Eye Foundation –
   San Antonio, TX
   Refractive Update
   September 10, 2000
   Category 1, Hours: 4.0
- Medical Education Collaborative Dallas, TX
   New Advances in Ophthalmic Fluroquinolones
   October 21, 2000
   Category 1, Hours: 1.5
- The University of Texas Houston Medical School Houston, TX
   Vision 2001 Spring Meeting
   March 24, 2001
   Category 1, Hours: 8.0
- The University of Texas Health Science Center San Antonio, TX
   New Treatment Paradigms in the Management of Glaucoma
   May 18-19, 2001
   Category 1, Hours: 3.75
  - The University of Texas Southwestern Medical

School - Dallas, TX

Ophthalmology Update: 20<sup>th</sup> Anniversary Seminar

September 8, 2001 Category 1, Hours: 7.0

- SLACK, Inc. Dallas, TX
   Three Targets for Glaucoma Management:
   A New Approach
   April 13, 2002
   Category 1, Hours: 3.5
- The Delaney Foundation San Antonio, TX Advanced Excellence in LASIK May 5, 2002 Category 1, Hours: 5.0
- The University of Texas Southwestern Medical School – Dallas, TX
   Clinical Applications of Ocular Bloodflow in Glaucoma & Age-Related Macular Degeneration October 5, 2002
   Category 1, Hours: 4.5
- The University of Texas Medical Branch Galveston, TX
   Office of Continuing Education Medical Therapy of Glaucoma 2002: Prostoglandins and More October 10, 2002 Category 1, Hours: 1.0
- Seton HealthCare Network Austin, TX Brain & Spine Center at Brackenridge Current Concepts in Stroke November 16, 2002 Category 1, Hours: 7.0
- Primary Care Network, Inc. Houston, TX
   The Headache Patient: Practical Strategies for Diagnosis and Treatment
   November 23, 2002
   Category 1, Hours: 4.0
- Lumenis San Antonio, TX
   Selective Laser Trabeculoplasty:
   The Latest Advance in Glaucoma Therapy

November 21, 2002 Informal

St. David's Medical Center – Austin, TX
 St. David's Grand Rounds 2003:
 Documentation – First Line Malpractice Defense
 January 7, 2003
 Category 1, Hours: 1.0

Primary Care Network, Inc. – Austin, TX
 Asthma: A Comprehensive Approach to Detection
 & Management
 March 1, 2003
 Category 1, Hours: 4.0

The Dulaney Foundation – Austin, TX
 Ocular Allergy: New Concepts in Therapy
 March 20, 2003
 Category 1, Hours: 1.0

 Scott and White Memorial Hospital – Temple, TX Everett R. Veirs Lecture & Ophthalmology Conference April 26, 2003 Category 1, Hours: 7.0

 SLACK, Inc. – Las Vegas, NV 1<sup>st</sup> Annual Ocular Surgery News Symposium Glaucoma: Improving Your Odds June 6-7, 2003 Category 1, Hours: 11.0

 Texas Medical Liability Trust – Austin, TX Don't Make Me Sue You June 27, 2003 Category 1, Hours: 1.0 Ethics, Hours: 1.0

Boron Lepore
 Applying the Data to Contemporary Clinical
 Practice: Managing Elevated Intraocular Pressure
 June 30, 2003

 Informal, Hours: 1.0

 The Dulaney Foundation – Austin, TX Fluroquinolone Update

July 22, 2003

Category 1, Hours: 1.0

- National Association of Managed Care Physicians Immune Based Dry Eye: A Progressive Disease August 2003
   Category 1, Hours: 1.0
- The Dulaney Foundation San Antonio, TX
   New and Emerging Techniques & Technology in Cataract & Refractive Surgery
   September 13, 2003
   Category 1, Hours: 11.0
- The Dulaney Foundation Austin, TX Procedures for the Glaucoma Patient September 18, 2003 Category 1, Hours: 1.0
- Texas Medical Liability Trust Austin, TX
  Medical Errors, Mandatory Disclosure & You
  November 18, 2003
  Category 1, Hours: 3.0
  Ethics, Hours: 1.0
- VISX Austin, TX
   Physician CustomVue Certification Course
   November 23, 2003
   Certification
- Bausch & Lomb Surgical Austin, TX
  Technolas 217A Laser Training
  September 11, 2003
  Certification
- Primary Care Network Austin, TX
   Evidence-Based Medicine: A Framework for Clinical Practice
   February 7, 2004
   Category 1, Hours: 4.0
- American Medical Association Austin, TX Depression in Primary Care February 20, 2004 Informal, Hours: 1.0

- Texas Medical Association Austin, TX
  Defensive Documentation Austin
  February 24, 2004
  Category 1, Hours: 3.0
  Ethics, Hours: 3.0
- Alcon & The AOS Austin, TX Allergy/Dry Eye Update March 11, 2004 Informal, Hours: 2.0
- Texas Medical Association Austin, TX E&M Documentation March 16, 2004 Category 1, Hours: 3.0 Ethics, Hours: 1.0
- Pfizer Austin, TX
   Interactive Roundtable Discussion on the Management of Glaucoma
   March 31, 2004
   Informal, Hours: 1.0
- Alcon Laboratories, Inc. Naples, FL Glaucoma Advisory Summit April 2 – 4, 2004 Informal, Hours: 8.0
- Maryland Research Institute Cancun, Mexico
   Otsuka Dry Eye Study Coordination Conference
   PPD Development
   April 19 21, 2004
   Informal, Hours: 8.0
- The Dulaney Foundation Austin, TX
   Blue Light and IOL Designs
   April 26, 2004
   Category 1, Hours: 1.0
- Scott and White Memorial Hospital Temple, TX Everett R. Veirs Lecture & Ophthalmology Conference May 1, 2004 Category 1, Hours: 6.0

Texas Medical Association – Austin, TX
 TexMed 2004 – Ophthalmology Day 2
 May 15, 2004
 Category 1, Hours: 7.0
 Ethics, Hours: 3.0

Ophthalmology Update – Austin, TX
 Glaucoma Management: IOP Lowering Agents
 June 9, 2004
 Category 1, Hours: 1.0

University of Florida – Austin, TX
 The Emerging Role for Neuroprotection in the
 Management of Glaucomatous Optic Neuropathy
 June 15, 2004
 Category 1, Hours: 0.5

Novartis Ophthalmics – Austin, TX
 AMD: The Fight for Sight
 June 24, 2004
 Informal, Hours: 1.0

Allergan – Austin, TX
 Teleconference: Restasis
 July 21, 2004
 Informal, Hours: 1.0

 The Dulaney Foundation – Austin, TX LASIK Flap Complications: The next step in prevention and management July 22, 2004 Category 1, Hours: 1.0

Interactive Information Solutions – Austin, TX
 Corneal Wound Healing: A Review of ARVO
 2004 Abstracts
 July 29, 2004
 Category 1, Hours: 1.0

Inspire Pharmaceuticals – Austin, TX
 A New Multiaction Therapy for Itch Associated with Allergic Conjunctivitis
 August 12, 2004
 Informal, Hours: 1.0

- Alcon Laboratories, Inc. San Antonio, TX
   Ophthalmic Symposium: Advances in Anterior
   Segment Surgery
   August 28, 29, 2004
   Category 1, Hours: 4.0
- Postgraduate Institute for Medicine Austin, TX
   Cystoid Macular Edema: New Dynamics for
   Prophylaxis and Treatment
   September 8, 2004
   Category 1, Hours: 1.0
- Austin Ophthalmology Society Austin, TX
   Pfizer Ophthalmics
   Update on the Management of Glaucoma
   September 9, 2004
   Informal, Hours: 1.0
- The New York Eye and Ear Infirmary Institute for Continuing Medical Education—New Orleans, LA Winds of Change: A Evidence-Based Approach October 22, 2004 Category, 1, Hours: 1.5
- The New York Eye and Ear Infirmary Institute for Continuing Medical Education-New Orleans, LA Forge: Focusing Ophthalmology on Reframing Glaucoma Evaluation October 23, 2004 Category 1, Hours: 1.5
- The New York Eye and Ear Infirmary Institute for Continuing Medical Education-New Orleans, LA What's New in Retinal Imaging: What Every Comprehensive Ophthalmologist Needs to Know October 24, 2004 Category 1, Hours: 1.5
- VISX Austin, TX
   VISX Fourier Wavefront Upgrade a CustomVue
   Technology
   October 28, 2004
   Informal, Hours: 1.0

- Texas Medical Association Austin, TX
   Hallway Consultations & Professional Courtesy
   November 18, 2004
   Category 1, Hours: 3.0
   Ethics, Hours: 3.0
- The Dulaney Foundation Las Vegas, NV Refractive IOL Symposium December 4-5, 2004 Category 1, Hours: 11.0
- VISX Houston, TX
   CustomVue VISX Technology Update
   February 16, 2005
   Informal, Hours: 3.0
- American Academy of Ophthalmology and Texas Ophthalmology Association – Austin, TX CodeQuest Ophthalmic Coding College 2005: Coding, Documentation & Compliance Seminar March 5, 2005 Category 1, Hours: 6.0
- The Dulaney Foundation Austin, TX
   Glaucoma 2005
   March 10, 2005
   Category 1, Hours: 1.0
- Texas Health Research Institute Dallas, TX 27<sup>th</sup> Annual Spring Ophthalmology Symposium April 1, 2005
   Category 1, Hours: 7.0
- Neuroscience Dallas, TX
   Link between Neurotransmitters and Hormones
   April 2, 2005
   Category 1, Hours: 4.0
- The Dulaney Foundation Fort Worth, TX Apodized Diffractive Lens Symposium April 9, 2005
   Category 1, Hours: 5.0
- SLACK, Inc. Houston, TX
   Update on the Management of Diabetic
   Retinopathy and its Complications

April 16, 2005

Category 1, Hours: 4.0

- The Dulaney Foundation San Antonio, TX Allergy Update April 18, 2005 Category 1, Hours: 1.0
- Price Vision Group Indianapolis, IN Advanced Cornea Course April 26 & 27, 2005
   Category 1, Hours: 13.0
- National Association of Managed Care Physicians – Austin, TX
   Emerging Trends in the Successful Diagnosis and Treatment of Chronic Dry Eye Disease May 17, 2005
   Category 1, Hours: 1.0
- The Dulaney Foundation Dallas, TX
   Revolutions in Cataract Business & Marketing
   May 22, 2005
   Category 1, Hours: 3.0
- Advanced Medial Optics, Inc. Austin, TX ReZoom Multifocal IOL July 1, 2005
   Certification
- The Dulaney Foundation San Antonio, TX Ophthalmic Symposium August 26-28, 2005 Category 1, Hours: 7.5
- The Dulaney Foundation Austin, TX Allergy and Dry Eye Update September 15, 2005 Category 1, Hours: 1.0
- Scott and White Memorial Hospital Temple, TX Everett R. Veirs Lecture & Ophthalmology Conference October 1, 2005 Category 1, Hours: 7.0

- American Academy of Ophthalmology Chicago, IL AAO Conference: Subspecialty & Annual Meeting October 14-18, 2005
   Category 1, Hours: 17.0
- The Dulaney Foundation Chicago, IL Phaco and Refractive Pearls From Around the World October 15, 2005 Category 1, Hours: 3.0
- Optos Chicago, IL
   Optos Academy Workshop
   Informal, Hours: 1.5
- ASCRS Chicago, IL Redefining Lenticular Refractive Surgery October 17, 2005
   Category 1, Hours: 1.5
- Texas Medical Association Austin, TX Coordination of Care 2005 October 18, 2005 Category 1, Hours: 3.0 Ethics, Hours: 3.0
- Medical Education Collaborative Austin, TX Managing the Risk of Intravitreal Injections October 27, 2005 Category 1, Hours: 1.5
- Neuroscience San Antonio, TX
   Neurotransmitters and Adrenal Stress
   February 7, 2006
   Category 1, Hours: 5.0
- Allergan Houston, TX
   Dry Eye Speaker Bureau Update Meeting
   March 3-5, 2006
   Informal, Hours: 12.0
- ASCRS San Francisco, CA
   March 17-22, 2006
   Informal, Hours: 20.0
- Texas Health Resources Dallas, TX

The 28<sup>th</sup> Annual Spring Ophthalmology Symposium March 24, 2006 Category 1, Hours: 7.0

- Texas Medical Association Austin, TX Retina Case Conundrums May 25, 2006 Category 1, Hours: 1.0
- Neuroscience Dallas, TX
   Neurochemical and Hormonal Consequences of the Modern Lifestyle: Avenues to Overcome the Resulting Imbalances
   June 17, 2006
   Category 1, Hours: 7.0
- Center for Accredited Healthcare Education Austin, TX
   Retinopathy Reporter: An Expert Dialogue on Diabetic Retinopathy Spring 2006 Issue June 23, 2006
   Category 1, Hours: 0.75
- Neuroscience Austin, TX
   ADHD: Attention, Hyperactivity & the Adrenal Gland
   July 12, 2006
- Neuroscience Austin, TX
   PMS, Menopause and Dysmenorrhea:
   Looking Beyond Hormones
   July 26, 2006
- The Dulaney Foundation San Antonio, TX
   Advances in Anterior Segment & Refractive Surgery
   August 26 & 27, 2006
   Category 1, Hours: 11.0
- Hawaiian Eye 2007 Kauai, HI
   January 13-19, 2007
   Category 1, Hours: 34.5
- Texas Medical Association Austin, TX Verdict 2007
   March 8, 2007
   Category 1, Hours: 3.0

Ethics, Hours: 3.0

Texas Medical Association – Austin, TX
 Retina Case Conundrums III 2007
 April 12, 2007
 Category 1, Hours: 2.0

The Dulaney Foundation – Austin, TX
 Ocular Allergy: Treatment Goals and
 Therapeutic Evaluation
 April 19, 2007
 Category 1, Hours: 1.0

- The Dulaney Foundation Austin, TX Innovations in Glaucoma Therapy May 10, 2007 Category 1, Hours: 1.0
- Texas Medical Foundation Austin, TX Electronic Medical Records 2007 Austin May 16, 2007 Category 1, Hours: 3.0 Ethics, Hours: 1.0
- The New York Eye & Ear Infirmary Institute for Continuing Medical Education—New Orleans, LA Managing Concomitant Eye Diseases: Expert Views on Glaucoma November 9, 2007 Category 1, Hours: 1.50
- American Academy of Ophthalmology New Orleans, LA
   Subspecialty Day – Refractive Surgery November 9 & 10, 2007
   Category 1, Hours: 14.0
- American Academy of Ophthalmology New Orleans, LA Annual Meeting November 10 – 13, 2007 Category 1, Hours: 9.0
- Texas Medical Association Austin, TX
   Ocular Emergencies
   January 10, 2008

Category 1, Hours: 2.0

- University of Kentucky MedEDirect Austin, TX NSAID Therapy from a Retinal Perspective February 21, 2008 Category 1, Hours: 1.0
- IntraLase Technology Austin, TX
   Physician Certification Program on IntraLase Technology
   March 3, 2008
   Certification
- University of Kentucky Austin, TX
   Glaucoma Therapy and the Ocular Surface
   March 27, 2008
   Category 1, Hours: 1.0
- Texas Health Resources Dallas, TX 30<sup>th</sup> Annual Spring Ophthalmology Symposium April 18, 2008 Category 1, Hours: 6.5
- University of Kentucky Austin, TX
   Ocular Allergy Learnings
   April 17, 2008
   Category 1, Hours: 1.0
- UT Southwestern Alumni Reunion Dallas, TX
   Science and Faith
   April 26, 2008
   Category 1, Hours: 1.0
- Texas Medical Association Austin, TX
   Retina Case Conundrums 2008,
   Current Concepts in ROP
   May 8, 2008
   Category 1, Hours: 2.0
- Texas Medical Association Austin, TX
   Promoting Physicians' Personal & Professional Fulfillment
   May 22, 2008
   Ethics, Hours: 1.0
- American Academy of Ophthalmology

   Atlanta, GA

2008 Subspecialty Day – Refractive Surgery November 7 & 8, 2008 Category 1, Hours: 14.0

- American Academy of Ophthalmology- Atlanta, GA 2008 Joint Meeting November 8-11, 2008 Category 1, Hours: 13.0
- Endo Optiks, Inc. Austin, TX
   Endoscopic Cyclophotocoagulation using the
   E2 Compact Microprobe™ Laser Endoscopy System
   May 19, 2009
   Certification
- Chylack, Inc. Austin, TX
   Lens Opacities Classification System Version III
   (LOCS III)
   August 1, 2009
   Certification
- National Retina Institute San Antonio, TX
   Ophthalmic Symposium
   August 28-30, 2009
   Category 1, Hours: 11.0
- American Academy of Ophthalmology –
   San Francisco, CA
   2009 Joint Meeting
   October 24-27, 2009
   Category 1, Hours: 10.0
- The Dulaney Foundation San Francisco, CA
   Prime Time CME Symposium
   October 25, 2009
   Category 1, Hours: 2.0
- The New York Eye And Ear Infirmary
   Institute for Continuing Medical Education
   San Francisco, CA
   Solving Diagnostic and Treatment Dilemmas with
   New Options for Ocular Infection and Inflammatory
   Conditions
   October 26, 2009
   Category 1, Hours: 1.5

- Lucentis RVO Program Austin, Texas
   July 22, 2010
   Informal Hours: 1.0 hour
- Ophthalmic Symposium San Antonio, Texas August 27-29, 2010
   Category 1, Hours: 11.0
- National Institutes of Health (NIH)
   Office of Extramural Research
   Protecting Human Research Participants
   September 7, 2010
   Certificate Number: 253583
- American Academy of Ophthalmology Chicago, IL
   2010 AAO Annual Meeting January 15, 2011 Category 1, Hours: 12.0
- American Academy of Ophthalmology Chicago, IL
   Subspecialty Day: Refractive Surgery January 15, 2011
   Category 1, Hours: 12.0
- American Society of Cataract and Refractive Surgery –
  San Diego, CA
   Eyeworld CME Educational Symposia
   Ethics of the Premium Channel
   March 27, 2011
   Category 1, Hours: 1.0
- Ophthalmic Symposium San Antonio, Texas August 27-28, 2011 Category 1, Hours: 11.5
- University of California School of Medicine San Francisco, California UCSF Glaucoma Update 2011 September 23 – 24, 2011 Category 1, Hours: 14.25
- Texas Medical Association Austin, Texas
  Beyond the White Coat: Physicians and Their
  Loved Ones
  October 4, 2011
  Category 1, Hours 1.0
- Hawaiian Eye 2012 Wailea, Maui Vindico Medical Education Taming Inflammation on the Ocular Surface: A Closer Look at Dry Eye. January 15, 2012 Category 1, Hours 1.0
- Hawaiian Eye 2012 Wailea, Maui Vindico Medical Education
   Practice Management: The Business of Ophthalmology January 15, 2012
   Category 1, Hours 1.5
- Hawaiian Eye 2012 Wailea, Maui Vindico Medical Education Cataract/IOL January 16, 2012 Category 1, Hours 4.0
- Hawaiian Eye 2012 Wailea, Maui Vindico Medical Education Cataract Surgery Complications; Mini Symposium on Femtosecond-Assisted Phacoemulsification; and Panel Discussion: Refractive Surgery Complications. January 17, 2012 Category 1, Hours 4.0
- Hawaiian Eye 2012 Wailea, Maui Vindico Medical Education Glaucoma January 18, 2012 Category 1, Hours 4.0
- Hawaiian Eye 2012 Wailea, Maui Vindico Medical Education
   Current Perspectives on the Optimal Management of Postsurgical Ocular Inflammation
   January 18, 2012

- Category 1, Hours 1.0
   Hawaiian Eye 2012 Wailea, Maui
   Specialty Symposium: Medical Retina Update for the
   Comprehensive Ophthalmologist; Management of the
   Ocular Surface, Part 1; and Management of the Ocular
   Surface, Part 2.
   January 19, 2012
   Category 1, Hours 4.0
- Hawaiian Eye 2012 Wailea, Maui
  Best Practices for Optimizing Postsurgical Outcomes
  January 19, 2012
  Category 1, Hours 1.0
- PPD Sunovion Training Austin, Texas
   Protocol review, highlights, Ophthalmic key points,
   Logistics and training.
   August 28, 2012
   Informal: 1 hour
- Texas Medical Association Austin, Texas International Ophthalmology October 23, 2012 Ethics, Hours 1.0
- American Academy of Ophthalmology Chicago, IL
   2012 AAO Annual Meeting November 9 – 13, 2012 Category 1, Hours: 20.0
- ACES/SEE Caribbean Eye Meeting San Juan, PR February 8 – 12, 2013
   Category 1, Hours: 17.0
- Glaukos® Austin, Tx
   April 15, 2013
   Glaukos® Physcian Training Program
   Glaukos iStent® Trabecular Micro-Bypass Stent
   Certificate of Completion
- Ophthalmic Symposium San Antonio, Tx August 24-25, 2013
   Category 1 Hours: 11.5

Thomas Henderson, M.D., F.A.C.S.

09/19/16

Date

#### **TEXAS MEDICAL BOARD**

P.O. BOX 2029 • AUSTIN, TEXAS 78768-2029

PHYSICIAN FULL PERMIT

LICENSE/PERMIT NUMBER F4863

THOMAS THOMAN HENDERSON, MD 3410 FAR WEST BLVD STE 140 AUSTIN TX 78731-3167 EXPIRATION DATE 08/31/2019

THIS CERTIFIES THAT THE LICENSEE/PERMIT HOLDER NAMED AND NUMBERED HEREON HAS PROVIDED THIS BOARD THE INFORMATION REQUIRED AND HAS PAID THE FEE FOR REGISTRATION FOR THE PERIOD INDICATED ABOVE PLEASE KEEP THIS BOARD NOTIFIED OF CHANGE OF ADDRESS



The National Institutes of Health (NIH) Office of Extramural Research certifies that **Thomas Henderson** successfully completed the NIH Web-based training course "Protecting Human Research Participants".

Date of completion: 09/10/2016.

Certification Number: 1786606.

### VALERIE E. GATAVASKI, COA 9100 WATERFORD CENTRE BOULEVARD #271 AUSTIN TX. 78758 (860)861-4470, vewash@yahoo.com

#### **PROFILE**

Well organized and proficient at multitasking. Extremely detail oriented and focused. Highly effective verbal and written communication skills. Maintain professionalism while working with patients in an empathetic and caring manner. Easy to work with; a cooperative and supportive team player.

#### **CAREER HIGHLIGHTS**

EYE CLINIC OF AUSTIN, Austin TX Certified Ophthalmic Assistant Research/Study Coordinator 2015 to Present

- Preliminary and ancillary testing includes the use of manual/automated lensometry.
- EHR/EDC documentation of all patient/subject histories, performed and recorded visual acuity.
- Proficient at pupil assessment, manual refraction with the use of phoropter, trial frame and lenses.
- Proficient in the use of Humphrey Visual Field Analyzer, Optical Coherence Tomography and Optos.
- Proficient in the assessment of intraocular pressure by means of Goldmann, Tonopen and Perkins devices.
- Proficient with EDC entries, maintaining all subject study binders, handling /shipping of specimens.
- Proficient in filing reports to a central or local IRB per study.
- Protocol, Informed Consent construction, current GCP, NIH, IATA certificates

### MIDDLESEX EYE PHYSICIANS, Middletown, CT

2012 to 2015

Certified Ophthalmic Assistant

- Preliminary testing, patient histories, assessment of visual acuity, manual refractions and assessment of intraocular pressure.
- Ascan, ultrasound biometry, acquired corneal curvature, axial length, anterior chamber depth using the IOL Master, Lenstar, Verion, manual Ascan with immersion, manual keratometry.
- Corneal assessment using Zeiss Corneal Topographer.

### THE EYE CARE GROUP, New Haven CT

2001 to 2012

Ophthalmic Assistant/Surgery Coordinator

- Met with patients, scheduled all appointments for surgical procedures, prepared necessary paperwork
- Scheduled and followed up on all ancillary testing prior to procedures.
- Acquired any necessary authorization/pre-certification from insurance carriers.

- Counseled patients with regard to proposed procedures, including the use of pre/post operative medication and restrictions. Informed the surgeons of schedules including revisions, routing all charts to the surgeons in a timely manner prior to the day of surgery
- Informed the surgeons of schedules including revisions, routing all charts to the surgeons in a timely manner prior to the day of surgery.

#### **EDUCATION**

National Institutes of Health - Good Clinical Practice and Protection of Human Research Subjects

JCAHPO Certification - Certified Ophthalmic Assistant

Stone Academy, Hamden CT – Medical Assisting

Wilbur L Cross High School, New Haven, CT – Diploma

#### **ORGANIZATIONS**

ASSOCIATION OF CLINICAL RESEARCH PROFESSIONALS
MEMBER 2016
SOCIETY OF CLINICAL RESEARCH ASSOCIATES
MEMBER 2017

cypdated 10-18-14 Value & Datavaski, COA.

# JOINT COMMISSION ON ALLIED HEALTH PERSONNEL IN OPHTHALMOLOGY® 2025 Woodlane Drive • St. Paul, Minnesota 55125-2998 PHONE (651) 731-2944 • (800) 284-3937 • FAX (651) 731-0410

#### **CERTIFICATION I.D.**

NAME

Valerie E. Gatavaski

I.D.#

209805

CERTIFICATION LEVEL

COA

EXPIRATION DATE

December 31, 2019



Clinical Research Education/Professional Certification

Valerie E. Gatavaski Member ID 60486 Member through 8/1/2018

MEMBERSHIP CARD www.socra.org

#### BASIC LIFE SUPPORT

## Provider



VALERIE E. GATAVASKI

The above individual has successfully completed the cognitive and skills evaluations in accordance with the curriculum of the American Heart Association Basic Life Support (CPR and AED) Program.

BASIC LIFE SUPPORT

Training

Center Name A-TCEMS TC ID#

TX04794

TC

Info Austin, TX 78721

512-978-0100

Course

Location

3410 Far West Blvd. Ste 140

Instructor Name

Sherry P. Hamilton

inst ID # 03130159373

Holder's Signature

Tampering with this card will alter its appearance. 15-1805



| PI/SITE NAIVIE: | | | | | |
|---|---|---|---|---|---|
| SUBJECT NAME: | | | | | |
| | DOCUMENTING THE CONSEN | T PROCESS | | | |
| Date: | | | | | |
| Consent Forms (CFs) r ☐ Main Study | reviewed:<br>CF, Version/Date: | | _ | | |
| Language of CF(s) revie | ewed: | | | | |
| Study Staff Member(s) | ☐ Spanish ☐ Other, Specify: Conducting CF discussion: | | | | |
| Was time allowed to as | | □ Vos | CD N - | | ₩ |
| Was a copy of the signe | ed CF(s) provided to the study subject? xplain: | □ Vaa | | | - |
| Was/were the CF(s) sig | ned prior to initiation of study procedures?<br>xplain: | □ Yes | □ No | | - |
| Additional Notes: | | | æ | | - |
| 3 | | | | | |
| i, | | | | | |
| | 2 | | | | |
| | | | | | L |
| | aining consent Date | | | a<br>24 | |

NON-REPORTABLE EVENT FORM (SUBMISSION OF INFORMATION THAT SALUS IRB DOES NOT REQUIRE TO BE REPORTED)

2111 West Braker Lane, Suite 400 ● Austin, TX 78758 ● P: 512.380.1244 ● F: 512.382.8902 ● <u>salus@salusirb.com</u>

SPONSOR: GUARDION HEALTH SCIENCES PROTOCOL#: 1 VERSION Z 77DEC ZOIS

INVESTIGATOR NAME: THOMAS HENDERSON, MAI)

#### A. REPORTING GUIDELINES:

If you are not familiar with Salus IRB reporting requirements regarding unanticipated problems (UPs), deviations, and other safety information, refer to the guidance document, "Reporting Guidelines For Unanticipated Problems, Deviations, and Other Safety Information," on the Salus IRB website.

Reports that must be submitted are those reports that indicate a new or increased risk of harm to research participants or others. Generally, to be reportable such an event should be unknown to the IRB and requires an action taken to minimize the risk to participants. For example, a safety-related change to the protocol, additional disclosure of risk in the consent form or IB, or other corrective action.

If you are required by your site or sponsor policy to submit IND Safety, MedWatch, SUSAR, or CIOMS Reports, or other safety information that does not meet the definition of an unanticipated problem and, therefore, does not require reporting to Salus IRB, use this form.

Salus IRB does not require reporting of minor protocol deviations. If you are required by your site or sponsor policy to submit minor protocol deviations, use this form.

For those events that Salus IRB does not require to be reported, if in the PI's judgment, any adverse events, minor protocol deviations or other events, when considered together indicate that changes to the research plan and/or consent form should be made, then the PI should provide an analysis of the events and any rationale for suggested changes at the time of continuing review, interim review, and/or site closure.

#### B. REPORT TYPE:

1. Minor Unplanned Protocol Deviation — is defined as an accidental or unintentional deviation from the Salus IRB-approved protocol that did not involve a new or increased risk to one or more research participants, did not adversely affect the rights, safety, or welfare of one or more participants, and did not adversely affect the conduct of the study.

Examples are: participant missed visit due to holidays, participant failed to return diary, participant failed to initial every page of the consent form, or other deviations that involve only logistical issues or only affect administrative aspects of the study.

a. Describe deviation or attach a description to this report (list each deviation being submitted by date of deviation and participant ID #):

OR

Subject 11921 R-ML DEVIATION DATE 11 JUL 2018 VISITS Subjects Visits. 7 WEEKS out of ININDOW DUE TO SCHEDULING CONFLICTS & Subject TRAVELLING ONT of THE AREA.

| EDONGOD GUI | HZZI IN HEALTH<br>SCIENCES | | | -7>- W |
|---|---|---|---|---|
| ii — | | PROTOCOL#: \ | VERSION Z | 27JEC 2014 |
| INVESTIGATOR | NAME: | LENDERSON, M. | 5 | |
| submitt | e Event, IND Safety, Meded to satisfy site or sporting ipated problem. | dWatch, SUSAR or CIOnsor reporting requiren | OMS Report, or nents, which doe | other safety information being<br>es not meet the criteria of ar |
| b.<br>OR | participant ID #): Report Type: | | illed by report | number, date of report, and |
| 3. Other ( | please describe): | | | |
| C. <u>INVESTIGAT</u> | OR OR SPONSOR REI | PRESENTATIVE STA | TEMENT: | |
| increased risks to pa<br>reporting of events w<br>report and attached de<br>review of this submi | s IRB requires only report rticipants or others. Furth hich do not meet the unanticuments to satisfy my site ssion and that Salus IRB very by signing this form, I ce | ing of events determined<br>er, I understand that bed<br>cipated problem criteria.<br>or sponsor requirements.<br>will only acknowledge re | d to be unanticipal cause of this policy of the policy of the policy of the policy of the policy of the policy of the policy of this submitted to the policy of the policy | t and the attached documents. In ated problems involving new or cy, Salus IRB does not require whedge that I am submitting this Salus IRB will not provide IRB mission. Further, if I am not the formation and sign this form on |
| Printed Name of Inve | T HENDERZ CON stigator/Authorized Designe | ee (Site) or Sponsor Repre | esentative (Sponso | or) |
| Signature of Investiga | THENDERSON<br>tor/Authorized Designee (S | ite) or Sponsor Represent | tative (Sponsor) | Date |
| SALUS IRB USE OF | NLY | | | |
| IRB STAFF ACKNO | OWLEDGEMENT OF RE | ECEIPT: | | |
| Irina H | nderson | y the IRB. This report ha | us been received an | nd filed in the IRB study file. |
| Printed Name of IRB | Administrative Staff MAUN | | | DI Oct 2018 |
| Signature of IRB Adn | inistrative Staff | | | Date |

NON-REPORTABLE EVENT FORM (SUBMISSION OF INFORMATION THAT SALUS IRB DOES NOT REQUIRE TO BE REPORTED)

2111 West Braker Lane, Suite 400 ● Austin, TX 78758 ● P: 512.380.1244 ● F: 512.382.8902 ● <u>salus@salusirb.com</u>

SPONSOR. GUARDION HEALTH SCIENCES PROTOCOL#: | VEZSION Z ZZDEL ZOIZ INVESTIGATOR NAME: THOMAS HENDEZSON, W.D.

#### A. REPORTING GUIDELINES:

If you are not familiar with Salus IRB reporting requirements regarding unanticipated problems (UPs), deviations, and other safety information, refer to the guidance document, "Reporting Guidelines For Unanticipated Problems, Deviations, and Other Safety Information," on the Salus IRB website.

Reports that must be submitted are those reports that indicate a new or increased risk of harm to research participants or others. Generally, to be reportable such an event should be unknown to the IRB and requires an action taken to minimize the risk to participants. For example, a safety-related change to the protocol, additional disclosure of risk in the consent form or IB, or other corrective action.

If you are required by your site or sponsor policy to submit IND Safety, MedWatch, SUSAR, or CIOMS Reports, or other safety information that does not meet the definition of an unanticipated problem and, therefore, does not require reporting to Salus IRB, use this form.

Salus IRB does not require reporting of minor protocol deviations. If you are required by your site or sponsor policy to submit minor protocol deviations, use this form.

For those events that Salus IRB does not require to be reported, if in the PI's judgment, any adverse events, minor protocol deviations or other events, when considered together indicate that changes to the research plan and/or consent form should be made, then the PI should provide an analysis of the events and any rationale for suggested changes at the time of continuing review, interim review, and/or site closure.

#### B. REPORT TYPE:

1. Minor Unplanned Protocol Deviation — is defined as an accidental or unintentional deviation from the Salus IRB-approved protocol that did not involve a new or increased risk to one or more research participants, did not adversely affect the rights, safety, or welfare of one or more participants, and did not adversely affect the conduct of the study.

Examples are: participant missed visit due to holidays, participant failed to return diary, participant failed to initial every page of the consent form, or other deviations that involve only logistical issues or only affect administrative aspects of the study.

a. Describe deviation or attach a description to this report (list each deviation being submitted by date of deviation and participant ID #):

Subject 44-LBR DEVIATION DATE ZUTILLY 2018 VISITS.

Subjects VISIT 3 ZWEEKS ONLY WINDOW DUE TO AN

UNFORESEEM SCHEDWING CONFLICT ON BEHALF OF THE

Subject.

Form 320 Non-Reportable Event Form Version: 01March2014

| SPONSOR: | RDION HEALTH<br>SCIENCES | PROTOCOL#: \ VETZSION Z | 2705(2014 |
|---|---|---|---|
| INVESTIGATOR | NAME: | | |
| | 1 HONLAS | HENDERSON, IN). | |
| submit | se Event, IND Safety, Meted to satisfy site or specipated problem. | edWatch, SUSAR or CIOMS Report, or onsor reporting requirements, which do | other safety information being<br>ses not meet the criteria of ar |
| a.<br>b.<br><b>OR</b> | Report Identifier (list of participant ID #): Report Type: | each report being submitted by report | number, date of report, and |
| 3. | please describe): | | |
| C. INVESTIGA | TOR OR SPONSOR RE | PRESENTATIVE STATEMENT: | |
| increased risks to preporting of events we report and attached of review of this submarked in Principal Investigated the Principal Investigated Printed Name of Investigation of | articipants or others. Further the unant documents to satisfy my site ission and that Salus IRB or, by signing this form, I construct the satisfy my site ission and that Salus IRB or, by signing this form, I construct the satisfy my site ission and that Salus IRB or, by signing this form, I construct the satisfy my signing this form, I construct the satisfy my signing this form, I construct the satisfy my signing this form, I construct the satisfy my signing this form, I construct the satisfy my significant the satisfy my significant the satisfy my site is satisfy my site in the satisfy my site is satisfy my site in the satisfy my site is satisfy my site in the satisfy my site is satisfy my site in the satisfy my site is sati | rting of events determined to be unanticipe ther, I understand that because of this politicipated problem criteria. I therefore acknowled or sponsor requirements. I understand that will only acknowledge receipt of this subsertify that I am authorized to submit this in the energy of the sponsor Representative (Sponsor). Site) or Sponsor Representative (Sponsor) | pated problems involving new or icy, Salus IRB does not require owledge that I am submitting this at Salus IRB will not provide IRB mission. Further, if I am not the information and sign this form on |
| SALUS IRB USE O | | | |
| IRB STAFF ACKN | OWLEDGEMENT OF R | ECEIPT: | |
| Truna f | Administrative Staff Administrative Staff | by the IRB. This report has been received a | and filed in the IRB study file. Or Oct 2018 Date |

NON-REPORTABLE EVENT FORM

(SUBMISSION OF INFORMATION THAT SALUS IRB DOES NOT REQUIRE TO BE REPORTED)

2111 West Braker Lane, Suite 400 ● Austin, TX 78758 ● P: 512.380.1244 ● F: 512.382.8902 ● salus@salusirb.com

SPONSOR QUARDION HEALTH SCIENCES PROTOCOL#: 1 VETESION 2 127 DEC 2017

INVESTIGATOR NAME: THOMAS HEADERSON, M.D.

#### A. REPORTING GUIDELINES:

If you are not familiar with Salus IRB reporting requirements regarding unanticipated problems (UPs), deviations, and other safety information, refer to the guidance document, "Reporting Guidelines For Unanticipated Problems, Deviations, and Other Safety Information," on the Salus IRB website.

Reports that must be submitted are those reports that indicate a new or increased risk of harm to research participants or others. Generally, to be reportable such an event should be unknown to the IRB and requires an action taken to minimize the risk to participants. For example, a safety-related change to the protocol, additional disclosure of risk in the consent form or IB, or other corrective action.

If you are required by your site or sponsor policy to submit IND Safety, MedWatch, SUSAR, or CIOMS Reports, or other safety information that does not meet the definition of an unanticipated problem and, therefore, does not require reporting to Salus IRB, use this form.

Salus IRB does not require reporting of minor protocol deviations. If you are required by your site or sponsor policy to submit minor protocol deviations, use this form.

For those events that Salus IRB does not require to be reported, if in the PI's judgment, any adverse events, minor protocol deviations or other events, when considered together indicate that changes to the research plan and/or consent form should be made, then the PI should provide an analysis of the events and any rationale for suggested changes at the time of continuing review, interim review, and/or site closure.

#### В. **REPORT TYPE:**

Minor Unplanned Protocol Deviation – is defined as an accidental or unintentional deviation from the Salus IRB-approved protocol that did not involve a new or increased risk to one or more research participants, did not adversely affect the rights, safety, or welfare of one or more participants, and did not adversely affect the conduct of the study.

Examples are: participant missed visit due to holidays, participant failed to return diary, participant failed to initial every page of the consent form, or other deviations that involve only logistical issues or only affect administrative aspects of the study.

a. Describe deviation or attach a description to this report (list each deviation being submitted by date of deviation and participant ID #):

OR Subjects PCP INTERRIPTED USE of LUMERA & for ZWEEKS TO

RIO CAUSES of Subjects. MINIOR SPIKE IN BLOOD PRESSURE, LUMERA &

found noncontribution to ELEVATION of DUOD PRESSURE. ADDITIONAL

Hypertensive Medication Prescribed. Subjects Compliant Resumed

Form 320 Non-Reportable Event Form LUMERA &, A FOLLOW-UP TO THE PCP REVEALS A LUWERING

Version: 01March2014 of Subjects Tolodo Pressure.


| SPONSOR:<br>INVESTIGATOR | PROTOCOL#: | |
|---|---|---|
| submi | se Event, IND Safety, MedWatch, SUSAR or CIOMS Report, or ot tted to satisfy site or sponsor reporting requirements, which does cipated problem. | ther safety information being not meet the criteria of ar |
| a.<br>b. | Report Identifier (list each report being submitted by report n participant ID #): Report Type: Initial Follow-up # | umber, date of report, and |
| 3. Other | (please describe): | |
| C. INVESTIGA | TOR OR SPONSOR REPRESENTATIVE STATEMENT: | |
| increased risks to preporting of events report and attached review of this subm Principal Investigate the Principal Investigate Thomas | windicates that I have reviewed the information provided in this report a us IRB requires only reporting of events determined to be unanticipate participants or others. Further, I understand that because of this policy which do not meet the unanticipated problem criteria. I therefore acknowled documents to satisfy my site or sponsor requirements. I understand that Salus insistence and that Salus IRB will only acknowledge receipt of this submission, by signing this form, I certify that I am authorized to submit this inforgator's behalf. THEVERSON WD THERESON WD THERESO | ed problems involving new or<br>F, Salus IRB does not require<br>ledge that I am submitting this<br>alus IRB will not provide IRB<br>ssion. Further, if I am not the<br>rmation and sign this form on |
| SALUS IRB USE O | DNLY | |
| IRB STAFF ACK | NOWLEDGEMENT OF RECEIPT: | |
| Trina | his report was not reviewed by the IRB. This report has been received and | filed in the IRB study file. |
| Printed Name of IRE | 3 Administrative Staff | . () |
| Signature of IRB Ad | ministrative Staff | 01 Oct 2018 |
| Dignarme of IVD Wo | minionarive Statt | Date |

NON-REPORTABLE EVENT FORM (SUBMISSION OF INFORMATION THAT SALUS IRB DOES NOT REQUIRE TO BE REPORTED)

2111 West Braker Lane, Suite 400 ● Austin, TX 78758 ● P: 512.380.1244 ● F: 512.382.8902 ● salus@salusirb.com

SPONSOR: GUATEDION HEALTH SCIENCES

PROTOCOL#: | VERSION 2 ZTDE(ZVI)

INVESTIGATOR NAME: THOWAS HENDERSON, N.D.

#### A. REPORTING GUIDELINES:

If you are not familiar with Salus IRB reporting requirements regarding unanticipated problems (UPs), deviations, and other safety information, refer to the guidance document, "Reporting Guidelines For Unanticipated Problems, Deviations, and Other Safety Information," on the Salus IRB website.

Reports that must be submitted are those reports that indicate a new or increased risk of harm to research participants or others. Generally, to be reportable such an event should be unknown to the IRB and requires an action taken to minimize the risk to participants. For example, a safety-related change to the protocol, additional disclosure of risk in the consent form or IB, or other corrective action.

If you are required by your site or sponsor policy to submit IND Safety, MedWatch, SUSAR, or CIOMS Reports, or other safety information that does not meet the definition of an unanticipated problem and, therefore, does not require reporting to Salus IRB, use this form.

Salus IRB does not require reporting of minor protocol deviations. If you are required by your site or sponsor policy to submit minor protocol deviations, use this form.

For those events that Salus IRB does not require to be reported, if in the PI's judgment, any adverse events, minor protocol deviations or other events, when considered together indicate that changes to the research plan and/or consent form should be made, then the PI should provide an analysis of the events and any rationale for suggested changes at the time of continuing review, interim review, and/or site closure.

#### B. <u>REPORT TYPE</u>:

Minor Unplanned Protocol Deviation – is defined as an accidental or unintentional deviation from the Salus IRB-approved protocol that did not involve a new or increased risk to one or more research participants, did not adversely affect the rights, safety, or welfare of one or more participants, and did not adversely affect the conduct of the study.

Examples are: participant missed visit due to holidays, participant failed to return diary, participant failed to initial every page of the consent form, or other deviations that involve only logistical issues or only affect administrative aspects of the study.

a. Describe deviation or attach a description to this report (list each deviation being submitted by date of deviation and participant ID #):

Subject 18819 TJF. DEVIATION DATE 30 MAY 2018 VISITS.
Subjects Visit 3 3 WEEKS out of WINDOW SECONDARY TO
SCHEDULING CONFLICTS ON BEHALF of the Subject of TRAVELLING
OUT of the AREA.

| SPONSOR: GUAZDION HEALTH PROTOCOL#: 1 VERSION 2 27DEL ZOIT |
|---|
| INVESTIGATOR NAME: THOMAS HENDERSON, M.D. |
| I HOWAD HENDERSON, M.J. |
| 2. Adverse Event, IND Safety, MedWatch, SUSAR or CIOMS Report, or other safety information bein submitted to satisfy site or sponsor reporting requirements, which does not meet the criteria of a unanticipated problem. |
| <ul> <li>a. Report Identifier (list each report being submitted by report number, date of report, and participant ID #):</li> <li>b. Report Type:</li></ul> |
| 3. Other (please describe): |
| C. INVESTIGATOR OR SPONSOR REPRESENTATIVE STATEMENT: |
| My signature below indicates that I have reviewed the information provided in this report and the attached documents. understand that Salus IRB requires only reporting of events determined to be unanticipated problems involving new or increased risks to participants or others. Further, I understand that because of this policy, Salus IRB does not require reporting of events which do not meet the unanticipated problem criteria. I therefore acknowledge that I am submitting this report and attached documents to satisfy my site or sponsor requirements. I understand that Salus IRB will not provide IRE review of this submission and that Salus IRB will only acknowledge receipt of this submission. Further, if I am not the Principal Investigator, by signing this form, I certify that I am authorized to submit this information and sign this form or the Principal Investigator's behalf. THOMAS THENDERSON MD Printed Name of Investigator/Authorized Designee (Site) or Sponsor Representative (Sponsor) Signature of Investigator/Authorized Designee (Site) or Sponsor Representative (Sponsor) Date |
| SALUS IRB USE ONLY |
| IRB STAFF ACKNOWLEDGEMENT OF RECEIPT: |
| The information in this report was not reviewed by the IRB. This report has been received and filed in the IRB study file. Printed Name of IRB Administrative Staff |
| Signature of IRB Administrative Staff Date OI Oct Jo18 |
| Data Data |

NON-REPORTABLE EVENT FORM (SUBMISSION OF INFORMATION THAT SALUS IRB DOES NOT REQUIRE TO BE REPORTED)

2111 West Braker Lane, Suite 400 • Austin, TX 78758 • P: 512.380.1244 • F: 512.382.8902 • salus@salusirb.com

SPONSOR: GUARDION HEALTH PROTOCOL#: 1 VERSION 7 27 DEL 2017 INVESTIGATOR NAME: THEMAS HENDERSON, MIS).

#### A. REPORTING GUIDELINES:

If you are not familiar with Salus IRB reporting requirements regarding unanticipated problems (UPs), deviations, and other safety information, refer to the guidance document, "Reporting Guidelines For Unanticipated Problems, Deviations, and Other Safety Information," on the Salus IRB website.

Reports that must be submitted are those reports that indicate a new or increased risk of harm to research participants or others. Generally, to be reportable such an event should be unknown to the IRB and requires an action taken to minimize the risk to participants. For example, a safety-related change to the protocol, additional disclosure of risk in the consent form or IB, or other corrective action.

If you are required by your site or sponsor policy to submit IND Safety, MedWatch, SUSAR, or CIOMS Reports, or other safety information that does not meet the definition of an unanticipated problem and, therefore, does not require reporting to Salus IRB, use this form.

Salus IRB does not require reporting of minor protocol deviations. If you are required by your site or sponsor policy to submit minor protocol deviations, use this form.

For those events that Salus IRB does not require to be reported, if in the PI's judgment, any adverse events, minor protocol deviations or other events, when considered together indicate that changes to the research plan and/or consent form should be made, then the PI should provide an analysis of the events and any rationale for suggested changes at the time of continuing review, interim review, and/or site closure.

#### B. REPORT TYPE:

1. Minor Unplanned Protocol Deviation — is defined as an accidental or unintentional deviation from the Salus IRB-approved protocol that did not involve a new or increased risk to one or more research participants, did not adversely affect the rights, safety, or welfare of one or more participants, and did not adversely affect the conduct of the study.

Examples are: participant missed visit due to holidays, participant failed to return diary, participant failed to initial every page of the consent form, or other deviations that involve only logistical issues or only affect administrative aspects of the study.

a. Describe deviation or attach a description to this report (list each deviation being submitted by date of deviation and participant ID #):

Subject 4913 D-A DEVIDENM DATE 2 MAY 2018 VISIT 2

D. Subject interrupted use of Limean Ellumena Boost of 30 Days
Secondary to knee replacement surkery. Treduced use on June 1, 2018

D. HBOVE NAMED Subject - DEVIATION DATE 18 MAY 2018 VISITZ
Subjects Visitz II Days outed window secondary to Knee Surgery IN ABILITY to Drive & TRANSPORTATION ARRANGEMENTS MUST BE
Version: 01March2014

MADE TO KEEP Appointment.


| SPONSOR: GLIARDIUM HEALTH SCIENCES PROTOCOL#: 1 VERSION 2 27DEC 2014 |
|---|
| INVESTIGATOR NAME: |
| THOMAS HENDERSON, MD. |
| 2. Adverse Event, IND Safety, MedWatch, SUSAR or CIOMS Report, or other safety information being submitted to satisfy site or sponsor reporting requirements, which does not meet the criteria of an unanticipated problem. |
| <ul> <li>a. Report Identifier (list each report being submitted by report number, date of report, and participant ID #):</li> <li>b. Report Type:</li></ul> |
| 3. Other (please describe): |
| C. INVESTIGATOR OR SPONSOR REPRESENTATIVE STATEMENT: |
| My signature below indicates that I have reviewed the information provided in this report and the attached documents. understand that Salus IRB requires only reporting of events determined to be unanticipated problems involving new of increased risks to participants or others. Further, I understand that because of this policy, Salus IRB does not require reporting of events which do not meet the unanticipated problem criteria. I therefore acknowledge that I am submitting this report and attached documents to satisfy my site or sponsor requirements. I understand that Salus IRB will not provide IRE review of this submission and that Salus IRB will only acknowledge receipt of this submission. Further, if I am not the Principal Investigator, by signing this form, I certify that I am authorized to submit this information and sign this form or the Principal Investigator's behalf. THOMAS THEOREM MD Printed Name of Investigator/Authorized Designee (Site) or Sponsor Representative (Sponsor) Date Signature of Investigator/Authorized Designee (Site) or Sponsor Representative (Sponsor) Date |
| SALUS IRB USE ONLY |
| IRB STAFF ACKNOWLEDGEMENT OF RECEIPT: |
| The information in this report was not reviewed by the IRB. This report has been received and filed in the IRB study file. Illustrative Staff |
| Signature of IRB Administrative Staff Date |

NON-REPORTABLE EVENT FORM (SUBMISSION OF INFORMATION THAT SALUS IRB DOES NOT REQUIRE TO BE REPORTED)

2111 West Braker Lane, Suite 400 ● Austin, TX 78758 ● P: 512.380.1244 ● F: 512.382.8902 ● salus@salusirb.com

SPONSOR: GLEARDION HEALTH SCIENCES

PROTOCOL#: | VERSION 2 27DEL ZOIF

INVESTIGATOR NAME: THOMAS 4 ENDERSON, N. D.

#### A. REPORTING GUIDELINES:

If you are not familiar with Salus IRB reporting requirements regarding unanticipated problems (UPs), deviations, and other safety information, refer to the guidance document, "Reporting Guidelines For Unanticipated Problems, Deviations, and Other Safety Information," on the Salus IRB website.

Reports that must be submitted are those reports that indicate a new or increased risk of harm to research participants or others. Generally, to be reportable such an event should be unknown to the IRB and requires an action taken to minimize the risk to participants. For example, a safety-related change to the protocol, additional disclosure of risk in the consent form or IB, or other corrective action.

If you are required by your site or sponsor policy to submit IND Safety, MedWatch, SUSAR, or CIOMS Reports, or other safety information that does not meet the definition of an unanticipated problem and, therefore, does not require reporting to Salus IRB, use this form.

Salus IRB does not require reporting of minor protocol deviations. If you are required by your site or sponsor policy to submit minor protocol deviations, use this form.

For those events that Salus IRB does not require to be reported, if in the PI's judgment, any adverse events, minor protocol deviations or other events, when considered together indicate that changes to the research plan and/or consent form should be made, then the PI should provide an analysis of the events and any rationale for suggested changes at the time of continuing review, interim review, and/or site closure.

#### B. REPORT TYPE:

1. Minor Unplanned Protocol Deviation – is defined as an accidental or unintentional deviation from the Salus IRB-approved protocol that did not involve a new or increased risk to one or more research participants, did not adversely affect the rights, safety, or welfare of one or more participants, and did not adversely affect the conduct of the study.

Examples are: participant missed visit due to holidays, participant failed to return diary, participant failed to initial every page of the consent form, or other deviations that involve only logistical issues or only affect administrative aspects of the study.

a. Describe deviation or attach a description to this report (list each deviation being submitted by date of deviation and participant ID #):

OR

Subject 11039JAT DEVIATION DATE ZZFEJZOIS V.Z. Subject REPORTS- DECREASING LALMERA LTO 1/2 DOSE DAILY SECONDAMY TO GLASTRO INTESTINAL ISSUES STARTING BUJANZOIS. Subject DIAGNOSES WITH INTESTINAL PARASITES - CONTRACTED Upon Eating SEAFOOD WHILE ON VACATION. Subject. DEEN IN FORLOW up by PCP, INTESTINALISSUES ARE RESOLVING.

| SPONSOR: GUARDION HEALTH SCIENCES PROTOCOL#: VERSION 2 Z FOEC 2017 INVESTIGATOR NAME: THOMAS HENDERSON, W.D. |
|---|
| LHOWAS HENDERSONI, WIJ- |
| 2. Adverse Event, IND Safety, MedWatch, SUSAR or CIOMS Report, or other safety information being submitted to satisfy site or sponsor reporting requirements, which does not meet the criteria of an unanticipated problem. |
| <ul> <li>a. Report Identifier (list each report being submitted by report number, date of report, and participant ID #):</li> <li>b. Report Type:</li></ul> |
| 3. Other (please describe): |
| C. INVESTIGATOR OR SPONSOR REPRESENTATIVE STATEMENT: |
| My signature below indicates that I have reviewed the information provided in this report and the attached documents. I understand that Salus IRB requires only reporting of events determined to be unanticipated problems involving new or increased risks to participants or others. Further, I understand that because of this policy, Salus IRB does not require reporting of events which do not meet the unanticipated problem criteria. I therefore acknowledge that I am submitting this report and attached documents to satisfy my site or sponsor requirements. I understand that Salus IRB will not provide IRB review of this submission and that Salus IRB will only acknowledge receipt of this submission. Further, if I am not the Principal Investigator, by signing this form, I certify that I am authorized to submit this information and sign this form on the Principal Investigator's behalf. Themes Therefore were the unanticipated problems involving new or increased risks to participated problems involving new or increased risks to be unanticipated by al |
| Signature of Investigator/Authorized Designee (Site) or Sponsor Representative (Sponsor) Date |
| SALUS IRB USE ONLY |
| IRB STAFF ACKNOWLEDGEMENT OF RECEIPT: |
| The information in this report was not reviewed by the IRB. This report has been received and filed in the IRB study file. Printed Name of IRB Administrative Staff OIOCT 2018 |
| Signature of IRB Administrative Staff Date |

NON-REPORTABLE EVENT FORM (SUBMISSION OF INFORMATION THAT SALUS IRB DOES NOT REQUIRE TO BE

REPORTED)

2111 West Braker Lane, Suite 400 ● Austin, TX 78758 ● P: 512.380.1244 ● F: 512.382.8902 ● salus@salusirb.com

SPONSOR: GUARDIUM HEALTH PROTOCOL#: 1 VERSIUM Z 27 DEL 2017

INVESTIGATOR NAME: THOMAS HENDERSON, M.J.

#### A. REPORTING GUIDELINES:

If you are not familiar with Salus IRB reporting requirements regarding unanticipated problems (UPs), deviations, and other safety information, refer to the guidance document, "Reporting Guidelines For Unanticipated Problems, Deviations, and Other Safety Information," on the Salus IRB website.

Reports that must be submitted are those reports that indicate a new or increased risk of harm to research participants or others. Generally, to be reportable such an event should be unknown to the IRB and requires an action taken to minimize the risk to participants. For example, a safety-related change to the protocol, additional disclosure of risk in the consent form or IB, or other corrective action.

If you are required by your site or sponsor policy to submit IND Safety, MedWatch, SUSAR, or CIOMS Reports, or other safety information that does not meet the definition of an unanticipated problem and, therefore, does not require reporting to Salus IRB, use this form.

Salus IRB does not require reporting of minor protocol deviations. If you are required by your site or sponsor policy to submit minor protocol deviations, use this form.

For those events that Salus IRB does not require to be reported, if in the PI's judgment, any adverse events, minor protocol deviations or other events, when considered together indicate that changes to the research plan and/or consent form should be made, then the PI should provide an analysis of the events and any rationale for suggested changes at the time of continuing review, interim review, and/or site closure.

#### B. REPORT TYPE:

1. Minor Unplanned Protocol Deviation – is defined as an accidental or unintentional deviation from the Salus IRB-approved protocol that did not involve a new or increased risk to one or more research participants, did not adversely affect the rights, safety, or welfare of one or more participants, and did not adversely affect the conduct of the study.

Examples are: participant missed visit due to holidays, participant failed to return diary, participant failed to initial every page of the consent form, or other deviations that involve only logistical issues or only affect administrative aspects of the study.

a. Describe deviation or attach a description to this report (list each deviation being submitted by date of deviation and participant ID #):

Subject 11039 JAT DEVIATION DATE 25 Apr. 2018 VISITZ
Subject Treports-Intercupter What Lumera Z Jor Fdays.
SECONDARY TO THE USE of ANTIBIOTICS for CONTINUED CASTRULINESTIMAL PARABITES. Subject HAS BEEN GERMIN
FOLLOW UP BY PCP - ISSUES Appears REJOLUED 30 Apr. 2018.

Form 320 Non-Reportable Event Form Version: 01March2014

| | 270512017 |
|---|---|
| INVESTIGATOR NAME: | |
| INVESTIGATOR NAME: | |
| <ol> <li>Adverse Event, IND Safety, MedWatch, SUSAR or CIOMS Report, or o<br/>submitted to satisfy site or sponsor reporting requirements, which does<br/>unanticipated problem.</li> </ol> | ther safety information being not meet the criteria of an |
| <ul> <li>a. Report Identifier (list each report being submitted by report reparticipant ID #):</li> <li>b. Report Type:</li></ul> | number, date of report, and |
| 3. Other (please describe): | |
| C. INVESTIGATOR OR SPONSOR REPRESENTATIVE STATEMENT: | |
| My signature below indicates that I have reviewed the information provided in this report a understand that Salus IRB requires only reporting of events determined to be unanticipated increased risks to participants or others. Further, I understand that because of this policy reporting of events which do not meet the unanticipated problem criteria. I therefore acknow report and attached documents to satisfy my site or sponsor requirements. I understand that S review of this submission and that Salus IRB will only acknowledge receipt of this submit Principal Investigator, by signing this form, I certify that I am authorized to submit this info the Principal Investigator's behalf. THOMAS THEODERSON MD Printed Name of Investigator/Authorized Designee (Site) or Sponsor Representative (Sponsor) Signature of Investigator/Authorized Designee (Site) or Sponsor Representative (Sponsor) | ed problems involving new or<br>y, Salus IRB does not require<br>eledge that I am submitting this<br>salus IRB will not provide IRB<br>ssion. Further, if I am not the<br>promation and sign this form on |
| SALUS IRB USE ONLY | |
| The information in this report was not reviewed by the IRB. This report has been received and Printed Name of IRB Administrative Staff What Addition | |
| Signature of IRB Administrative Staff | Ol Oct 2018 |
| | Duit |

NON-REPORTABLE EVENT FORM (SUBMISSION OF INFORMATION THAT SALUS IRB DOES NOT REQUIRE TO BE REPORTED)

2111 West Braker Lane, Suite 400 ● Austin, TX 78758 ● P: 512.380.1244 ● F: 512.382.8902 ● salus@salusirb.com

SPONSOR: (SWARDION HEALTH SCIENTEPROTOCOL#: | VERSION 2 27-DELZOIT

INVESTIGATOR NAME: THOMAS HE NIDER SON, MID

#### A. REPORTING GUIDELINES:

If you are not familiar with Salus IRB reporting requirements regarding unanticipated problems (UPs), deviations, and other safety information, refer to the guidance document, "Reporting Guidelines For Unanticipated Problems, Deviations, and Other Safety Information," on the Salus IRB website.

Reports that must be submitted are those reports that indicate a new or increased risk of harm to research participants or others. Generally, to be reportable such an event should be unknown to the IRB and requires an action taken to minimize the risk to participants. For example, a safety-related change to the protocol, additional disclosure of risk in the consent form or IB, or other corrective action.

If you are required by your site or sponsor policy to submit IND Safety, MedWatch, SUSAR, or CIOMS Reports, or other safety information that does not meet the definition of an unanticipated problem and, therefore, does not require reporting to Salus IRB, use this form.

Salus IRB does not require reporting of minor protocol deviations. If you are required by your site or sponsor policy to submit minor protocol deviations, use this form.

For those events that Salus IRB does not require to be reported, if in the PI's judgment, any adverse events, minor protocol deviations or other events, when considered together indicate that changes to the research plan and/or consent form should be made, then the PI should provide an analysis of the events and any rationale for suggested changes at the time of continuing review, interim review, and/or site closure.

#### B. REPORT TYPE:

Minor Unplanned Protocol Deviation – is defined as an accidental or unintentional deviation from the Salus IRB-approved protocol that did not involve a new or increased risk to one or more research participants, did not adversely affect the rights, safety, or welfare of one or more participants, and did not adversely affect the conduct of the study.

Examples are: participant missed visit due to holidays, participant failed to return diary, participant failed to initial every page of the consent form, or other deviations that involve only logistical issues or only affect administrative aspects of the study.

a. Describe deviation or attach a description to this report (list each deviation being submitted by date of deviation and participant ID #):

Subjects Visit Z bweeks outof window secondary to HEALTH ISSUES DESIGNATION DATE 22 APR 2018

- Subject has missed unknown number of doses of Lumerate

Form 320 Non-Reportable Event Form Subject Admits to SHAZING DOSES 

INITH 8 POUSE.

| SPONSOR: GUARDION HEALTH SCIENCES PROTOCOL#: 1 VERSION Z 77: INVESTIGATOR NAME: [HOWAS HENDERSON] W.1) | )EC 2017 |
|---|---|
| THOMAS HENDERSON, M.) | |
| 2. Adverse Event, IND Safety, MedWatch, SUSAR or CIOMS Report, or other sa submitted to satisfy site or sponsor reporting requirements, which does not a unanticipated problem. | afety information being<br>neet the criteria of an |
| <ul> <li>a. Report Identifier (list each report being submitted by report number participant ID #):</li> <li>b. Report Type:</li></ul> | r, date of report, and |
| 3. Other (please describe): | |
| C. INVESTIGATOR OR SPONSOR REPRESENTATIVE STATEMENT: | |
| My signature below indicates that I have reviewed the information provided in this report and the understand that Salus IRB requires only reporting of events determined to be unanticipated profince increased risks to participants or others. Further, I understand that because of this policy, Salur reporting of events which do not meet the unanticipated problem criteria. I therefore acknowledge report and attached documents to satisfy my site or sponsor requirements. I understand that Salus IR review of this submission and that Salus IRB will only acknowledge receipt of this submission. Principal Investigator, by signing this form, I certify that I am authorized to submit this information the Principal Investigator's behalf. THOMAS THADELSON MD Printed Name of Investigator/Authorized Designee (Site) or Sponsor Representative (Sponsor) Thomas Thadleson MD Signature of Investigator/Authorized Designee (Site) as Sponsor Representative (Sponsor) | blems involving new or is IRB does not require that I am submitting this RB will not provide IRB Further, if I am not the on and sign this form on |
| Signature of Investigator/Authorized Designee (Site) or Sponsor Representative (Sponsor) | Date |
| SALUS IRB USE ONLY | |
| IRB STAFF ACKNOWLEDGEMENT OF RECEIPT: | |
| The information in this report was not reviewed by the IRB. This report has been received and filed in the IRB. This report has been received and the IRB. This report has | in the IRB study file. |
| | 01 Oct 2018 |
| Signature of IRB Administrative Staff | Date |

NON-REPORTABLE EVENT FORM (SUBMISSION OF INFORMATION THAT SALUS IRB DOES NOT REQUIRE TO BE REPORTED)

2111 West Braker Lane, Suite 400 ● Austin, TX 78758 ● P: 512.380.1244 ● F: 512.382.8902 ● salus@salusirb.com

SPONSOR GUARDION HEALTH PROTOCOL#: | VERSION 2 27 DECZOIT INVESTIGATOR NAME: THOMAS HENDERSON, WW.

#### A. REPORTING GUIDELINES:

If you are not familiar with Salus IRB reporting requirements regarding unanticipated problems (UPs), deviations, and other safety information, refer to the guidance document, "Reporting Guidelines For Unanticipated Problems, Deviations, and Other Safety Information," on the Salus IRB website.

Reports that must be submitted are those reports that indicate a new or increased risk of harm to research participants or others. Generally, to be reportable such an event should be unknown to the IRB and requires an action taken to minimize the risk to participants. For example, a safety-related change to the protocol, additional disclosure of risk in the consent form or IB, or other corrective action.

If you are required by your site or sponsor policy to submit IND Safety, MedWatch, SUSAR, or CIOMS Reports, or other safety information that does not meet the definition of an unanticipated problem and, therefore, does not require reporting to Salus IRB, use this form.

Salus IRB does not require reporting of minor protocol deviations. If you are required by your site or sponsor policy to submit minor protocol deviations, use this form.

For those events that Salus IRB does not require to be reported, if in the PI's judgment, any adverse events, minor protocol deviations or other events, when considered together indicate that changes to the research plan and/or consent form should be made, then the PI should provide an analysis of the events and any rationale for suggested changes at the time of continuing review, interim review, and/or site closure.

#### B. REPORT TYPE:

Minor Unplanned Protocol Deviation — is defined as an accidental or unintentional deviation from the Salus IRB-approved protocol that did not involve a new or increased risk to one or more research participants, did not adversely affect the rights, safety, or welfare of one or more participants, and did not adversely affect the conduct of the study.

Examples are: participant missed visit due to holidays, participant failed to return diary, participant failed to initial every page of the consent form, or other deviations that involve only logistical issues or only affect administrative aspects of the study.

a. Describe deviation or attach a description to this report (list each deviation being submitted by date of deviation and participant ID #):

OR Subject 1831 MT3 DEVIATION DATE YMAY 2018 VISITZ

OSubject NOT DILATED AT VISIT PER THE PI BECAUSE.

OJ (R) BELL'S PALSY, Subject TO BE DILATED AT VISIT3 I

PALSY IS RESOLUED 
O. ABOUT MANIED SUBJECT MUSIED DOUES DEV. DATE - 2 AUG 2018

VISIT3 - Subject MUSSED DOSES THEN DIC LUMERA K-SECONDARY

Form 320 Non-Reportable Event Form
Version: 01March2014

TO INITESTIMAL UPSET & LETHARCAY, Subject SEEN BY PCP

DIAG NOSED WITH HSV. FLARE UP - AS of 28 AUG 2018 HSV RESOLVED -

| SPONSOR: GWARDION HEALTH WESPROTOCOL#: 1 VERSION 2 27 DELZOIT |
|---|
| INVESTIGATOR NAME: THOMAS HEADERSON, MI) |
| 2. Adverse Event, IND Safety, MedWatch, SUSAR or CIOMS Report, or other safety information being submitted to satisfy site or sponsor reporting requirements, which does not meet the criteria of an unanticipated problem. |
| <ul> <li>a. Report Identifier (list each report being submitted by report number, date of report, and participant ID #):</li> <li>b. Report Type:</li></ul> |
| 3. Other (please describe): |
| C. INVESTIGATOR OR SPONSOR REPRESENTATIVE STATEMENT: |
| My signature below indicates that I have reviewed the information provided in this report and the attached documents. I understand that Salus IRB requires only reporting of events determined to be unanticipated problems involving new or increased risks to participants or others. Further, I understand that because of this policy, Salus IRB does not require reporting of events which do not meet the unanticipated problem criteria. I therefore acknowledge that I am submitting this report and attached documents to satisfy my site or sponsor requirements. I understand that Salus IRB will not provide IRB review of this submission and that Salus IRB will only acknowledge receipt of this submission. Further, if I am not the Principal Investigator, by signing this form, I certify that I am prized to submit this information and sign this form on the Principal Investigator's behalf. THOMAS THEODERSON MD Printed Name of Investigator/Authorized Designee (Site) or Sponsor Representative (Sponsor) Date Date |
| Signature of investigator/Authorized Designee (Site) or Sponsor Representative (Sponsor) Date |
| SALUS IRB USE ONLY |
| IRB STAFF ACKNOWLEDGEMENT OF RECEIPT: |
| The information in this report was not reviewed by the IRB. This report has been received and filed in the IRB study file. **THE INDICATE OF THE STATE OF THE ST |
| Printed Name of IRB Administrative Staff Of Oct 7010 |
| Signature of IRB Administrative Staff Date |

### Statistical Analysis Plan

At the end of the trail period, data will be collected by the Principal Investigator and analyzed by professional optical engineers at Western University of Health Sciences, Pomona CA. The data provided will only contain patient ID, age, and sex, without containing any identifying details about each participant. Data will be analyzed upon measurement quality, according to the respective manufacturer procedures, in each outcome measure. In the event which data is missing or incomplete, we will evaluate the appropriate measures to include the available information and consult with qualified professionals.

Preliminary and sub-analyses will be performed using the statistical programing software, SPSS Systems. The objective is to examine the distribution and potential relationships within data sets through standardized descriptive-numerical summaries. Statistical analysis strategies may include a mixed-design Analysis Of Variance (ANOVA) to examine the following outcome measures across the three time-points of data collection; including visual acuity, contrast sensitivity, dark adaptation recovery, and MPOD levels. A post hoc sub-analysis of paired sample t-test may be used (either Bonferroni correction or Tukey test) to evaluate the change in each outcome measure parameter, if needed, in respect to each treatment group. Additionally, each group-measurement may be separated and analyzed by eye; to evaluate inter-eye differences from each treatment. Results of the statistical analysis will be analyzed as group averages of each outcome measurement.